CLINICAL TRIAL: NCT03038100
Title: A Phase III, Multicenter, Randomized, Study of Atezolizumab Versus Placebo Administered in Combination With Paclitaxel, Carboplatin, and Bevacizumab to Patients With Newly-Diagnosed Stage III or Stage IV Ovarian, Fallopian Tube, or Primary Peritoneal Cancer
Brief Title: A Study of Atezolizumab Versus Placebo in Combination With Paclitaxel, Carboplatin, and Bevacizumab in Participants With Newly-Diagnosed Stage III or Stage IV Ovarian, Fallopian Tube, or Primary Peritoneal Cancer
Acronym: IMagyn050
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Collaborators: GOG Foundation (Network); European Network of Gynaecological Oncological Trial Groups (ENGOT) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: YO39523; 2016-003472-52 (EudraCT Number)
Record Dates: First submitted 2017-01-30; First posted 2017-01-31 (Estimated); Results first posted 2023-02-17 (Actual); Last update posted 2023-02-17 (Actual); Status verified 2023-02

CONDITIONS: Ovarian Cancer; Fallopian Tube Cancer; Peritoneal Neoplasms
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms; Peritoneal Neoplasms | interventions — Paclitaxel; Carboplatin; atezolizumab; Bevacizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab (Experimental): Participants in the primary tumor-reductive surgery group will receive paclitaxel, carboplatin, atezolizumab intravenous (IV) infusion on Day 1 of each 21-day cycle for a total of 6 cycles, and bevacizumab IV infusion starting with Cycle 2 for a total of 5 cycles, followed by maintenance therapy bevacizumab with atezolizumab for a total of 22 cycles of atezolizumab and 21 cycles of bevacizumab. Participants in the neoadjuvant therapy group will receive paclitaxel, carboplatin and atezolizumab for 6 cycles and bevacizumab for 4 cycles. Interval surgery will occur between cycles 3 and 4. Each cycle is 21 days long. After 6 cycles, participants will start maintenance therapy of bevacizumab and atezolizumab for additional 16 cycles.
  Interventions: Drug: Paclitaxel; Drug: Carboplatin; Drug: Atezolizumab; Drug: Bevacizumab
- Placebo With Paclitaxel, Carboplatin and Bevacizumab (Placebo Comparator): Participants in the primary tumor-reductive surgery group will receive paclitaxel, carboplatin, atezolizumab placebo IV infusion on Day 1 of each 21-day cycle for a total of 6 cycles, and bevacizumab IV infusion starting with Cycle 2 for a total of 5 cycles, followed by maintenance therapy bevacizumab with atezolizumab placebo for a total of 22 cycles of atezolizumab placebo and 21 cycles of bevacizumab. Participants in the neoadjuvant therapy group will receive paclitaxel, carboplatin and placebo for 6 cycles and bevacizumab for 4 cycles. Interval surgery will occur between cycles 3 and 4. Each cycle is 21 days long. After 6 cycles, participants will start maintenance therapy of bevacizumab and placebo for additional 16 cycles.
  Interventions: Drug: Paclitaxel; Drug: Carboplatin; Drug: Bevacizumab; Drug: Atezolizumab Placebo

INTERVENTIONS:
Drug: Paclitaxel — Paclitaxel 175 milligrams per square meter (mg/m^2) IV infusion on Day 1 of each 21-day cycle
Drug: Carboplatin — Carboplatin at a dose to achieve a target area under the curve (AUC) of 6 milligrams per milliliter*minute (mg/mL*min) on Day 1 of each 21-day cycle for a total of 6 cycles
Drug: Atezolizumab — Atezolizumab 1200 mg IV infusion on Day 1 of each 21-day cycle
  Arms: Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab
Drug: Bevacizumab — Bevacizumab 15 milligrams per kilogram (mg/kg) IV infusion as per the schedule specified in respective arms
Drug: Atezolizumab Placebo — Placebo matching to atezolizumab on Day 1 of each 21-day cycle
  Arms: Placebo With Paclitaxel, Carboplatin and Bevacizumab

SUMMARY:
This is a Phase III, global, double-blind, 2-arm randomized study designed to compare the efficacy and safety of atezolizumab + paclitaxel + carboplatin + bevacizumab versus placebo + paclitaxel + carboplatin + bevacizumab. Study participants will have Stage 3 or 4 ovarian cancer (OC), fallopian tube cancer (FTC), or primary peritoneal cancer (PPC) with macroscopic residual disease postoperatively (i.e., after primary tumor reductive surgery) or who will undergo neoadjuvant therapy followed by interval surgery.

ELIGIBILITY:
Inclusion Criteria:

* Participants receiving a histologic diagnosis of epithelial ovarian cancer (EOC), peritoneal primary carcinoma, or fallopian tube cancer
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2
* Life expectancy greater than (>) 12 weeks
* For participants who receive therapeutic anticoagulation: stable anticoagulant regimen
* Availability of a representative formalin-fixed, paraffin-embedded (FFPE) tumor specimen in paraffin blocks (preferred) or at least 20 unstained slides (for detailed tissue requirements at screening)

Exclusion Criteria:

* Received a current diagnosis of borderline epithelial ovarian tumor (formerly tumors of low malignant potential)
* Have recurrent invasive epithelial ovarian, fallopian tube, or primary peritoneal cancer that was treated only with surgery (example [e.g.], participants with Stage IA or Stage IB epithelial ovarian or fallopian tube cancers)
* Have non-epithelial ovarian tumors (e.g., germ cell tumors, sex cord stromal tumors)
* Received prior radiotherapy to any portion of the abdominal cavity or pelvis
* Received prior chemotherapy for any abdominal or pelvic tumor that include neoadjuvant chemotherapy (NACT) for ovarian, primary peritoneal or fallopian tube cancer
* Received any biological and/or targeted therapy (including but not limited to vaccines, antibodies, tyrosine kinase inhibitors) or hormonal therapy for management and/or treatment of epithelial ovarian or peritoneal primary cancer
* Have synchronous primary endometrial cancer
* Have a prior history of primary endometrial cancer, except: Stage IA cancer; superficial myometrial invasion, without lymphovascular invasion; grade less than (<) 3 or poorly differentiated subtypes, and this includes papillary serous, clear cell or other International Federation of Gynecological Oncologists (FIGO) Grade 3 lesions
* With the exception of non-melanoma skin cancer and other specific malignancies as noted above, other invasive malignancies with any evidence of other cancers present within the last 5 years or previous cancer treatment that contraindicates this protocol therapy
* Have a known hypersensitivity or allergy to biopharmaceutical agents produced in Chinese hamster ovary cells or any component of the atezolizumab and/or bevacizumab formulations
* Undergo major surgical procedure within 28 days prior to first bevacizumab dose, or anticipation of the need for a major surgical procedure during the course of the study except participants who receive NACT and will need interval surgery. This may include but is not limited to laparotomy.
* Have prior allogeneic bone marrow transplantation or solid organ transplant
* Have any other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results
* Have any approved or investigational anti-cancer therapy, including chemotherapy or hormonal therapy, with exceptions: Hormone-replacement therapy or oral contraceptives
* Are administered treatment with any other investigational agent or participation in another clinical study with anti-cancer therapeutic intent
* Have core biopsy or other minor surgical procedures within 7 days prior to the first dose of bevacizumab
* Have known sensitivity to any component of bevacizumab
* Have known sensitivity to any component of paclitaxel
* Current treatment with anti-viral therapy for hepatitis B virus (HBV)
* History of leptomeningeal disease

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1301 (Actual)
Dates: Start 2017-03-08 (Actual); Primary Completion 2022-02-08 (Actual); Study Completion 2022-08-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (268):
- United States (127):
  - St. Joseph'S Hospital & Medical Center, Phoenix, Arizona
  - Arizona Oncology Associates, PC - HAL, Scottsdale, Arizona
  - Arizona Oncology - HOPE Wilmot, Tucson, Arizona
  - Moores Cancer Center at UC San Diego Health, La Jolla, California
  - LAC + USC Medical Center, Los Angeles, California
  - UCLA - School of Medicine, Los Angeles, California
  - Kaiser Permanente - Oakland, Oakland, California
  - The Center for Cancer Prevention and Treatment at St.Joseph Hospital of Orange, Orange, California
  - UC Irvine Medical Center, Orange, California
  - Stanford University, Palo Alto, California
  - Kaiser Permanente - Sacramento, Roseville, California
  - Southern California Kaiser Permanente, San Diego, California
  - California Pacific Medical Center Research Institute, San Francisco, California
  - K. Permanente - San Fransisco, San Francisco, California
  - University of California San Francisco Cancer Center, San Francisco, California
  - Kaiser Permanente - Santa Clara, Santa Clara, California
  - Olive View/Ucla Medical Center, Sylmar, California
  - Kaiser Permanente - Walnut Creek, Walnut Creek, California
  - University of Colorado Hospital - Anschutz Cancer Pavilion, Aurora, Colorado
  - Danbury Hospital, Danbury, Connecticut
  - Eastern Connecticut Hematology and Oncology Associates; (ECHO), Norwich, Connecticut
  - Sylvester Comprehensive Cent., Miami, Florida
  - Miami Cancer Institute of Baptist Health, Inc., Miami, Florida
  - Sarasota Memorial Health Care System; Cancer Research Program, Sarasota, Florida
  - Women's Cancer Associates, St. Petersburg, Florida
  - Northside Hospital, Atlanta, Georgia
  - Northeast Georgia Medical Center; Oncology Research Dept-5C, Gainesville, Georgia
  - Women's Cancer Center, Honolulu, Hawaii
  - Rush University Medical Center, Chicago, Illinois
  - Univ of Chicago, Chicago, Illinois
  - Sudarshan K. Sharma, MD, Ltd., Hinsdale, Illinois
  - Parkview Research Center, Fort Wayne, Indiana
  - St.Vincent Health System; Gynecologic Oncology, Indianapolis, Indiana
  - University of Iowa Hospital & Clinic; Division of Hematology/Oncology, Iowa City, Iowa
  - University of Kentucky; Gynecologic Oncology, Lexington, Kansas
  - St. Elizabeth Edgewood; Cancer Care Center? for Account St. Elizabeth Edgewood, Edgewood, Kentucky
  - Woman's Hospital, Baton Rouge, Louisiana
  - Maine Medical Partners Women's Health; Gyn-Oncology, Scarborough, Maine
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Weinberg CA Inst Franklin Sq, Baltimore, Maryland
  - Frederick Health Hospital, Frederick, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - St. Joseph Mercy Hospital, Ann Arbor, Michigan
  - Karmanos Cancer Institute, Detroit, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Sanford Health Bemidji, Bemidji, Minnesota
  - University of Minnesota, Minneapolis, Minnesota
  - Metro-Minnesota Community Oncology Research Consortium, Saint Louis Park, Minnesota
  - Minnesota Oncology Hematology Woodbury, Woodbury, Minnesota
  - St. Dominic-Jackson Memorial Hospital, Jackson, Mississippi
  - Washington University School of Medicine; Dept of Medicine/Div of Medical Oncology, St Louis, Missouri
  - Billings Clinic; Cancer Center, Billings, Montana
  - Community Cancer Care, Missoula, Montana
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Women's Cancer Center, Las Vegas, Nevada
  - Center of Hope, Reno, Nevada
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - MSK @Basking Ridge, Basking Ridge, New Jersey
  - Cooper Health System; MD Anderson Cancer Center, Camden, New Jersey
  - John Theurer Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey
  - Memorial Sloan Kettering Cancer Center; MSK Monmouth, Middletown, New Jersey
  - Jersey Shore Med Ctr; OB/GYN, Neptune City, New Jersey
  - Holy Name Hospital, Teaneck, New Jersey
  - Southwest Gynecologic Oncology Associates, Inc., Albuquerque, New Mexico
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Womens Cancer Care Association, Albany, New York
  - New York Presbyterian Queens, Flushing, New York
  - Northwell Health; Monter Cancer Center, Lake Success, New York
  - New York Univ Medical Center; Obstetrics & Gynecolog, New York, New York
  - Mount Sinai Downtown Chelsea Centre, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan-Kettering CC, Rockville Centre, New York
  - Levine Cancer Institute, Charlotte, North Carolina
  - Novant Health Presbyterain Medical Center, Charlotte, North Carolina
  - Duke Medical Center, Durham, North Carolina
  - Forsythe Memorial Hospital Inc., dba Novant Health Oncology Specialists, Winston-Salem, North Carolina
  - Wake Forest Baptist Medical Center, Winston-Salem, North Carolina
  - Sanford Health Bismarck, Bismarck, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - University of Cincinnati, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Univ Hospitals of Cleveland, Cleveland, Ohio
  - Fairview Hospital; Cleveland Clinic Cancer Center, Cleveland, Ohio
  - Columbus NCORP, Columbus, Ohio
  - Ohio State University, Arthur James Cancer Hospital, Columbus, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - University of Oklahoma; Stephenson Oklahoma Canc Ctr, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute, Tulsa, Oklahoma
  - Oncology Associates of Oregon, P.C.; Willamette Valley Cancer Institute, Springfield, Oregon
  - Northwest Cancer Specialists, P.C., Tigard, Oregon
  - University of Pennsylvania Health System; Cancer Center, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Magee-Woman's Hospital, Pittsburgh, Pennsylvania
  - Western Pennsylvania Hospital, Pittsburgh, Pennsylvania
  - Abington Mem Hosp-Abington; Rose. Can Ctr,Gyn Onc Ins, Willow Grove, Pennsylvania
  - WellSpan Gynecologic Oncology, York, Pennsylvania
  - Women & Infants Hospital, Providence, Rhode Island
  - Bon Secours - St. Francis Hospital, Greenville, South Carolina
  - Monument Health Rapid City Hospital, Inc., Rapid City, South Dakota
  - Sanford Health System, Sioux Falls, South Dakota
  - Dell Seton Medical Center at UT-Seton Infusion Center; Research Department, Austin, Texas
  - Texas Oncology Cancer Center, Austin, Texas
  - Texas Oncology, Bedford, Texas
  - UT Southwestern Medical Center at Dallas; Department of Pathology, Dallas, Texas
  - Texas Oncology, P.A. - Fort Worth, Fort Worth, Texas
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Houston Methodist Hospital, Houston, Texas
  - Rocky Mountain Cancer Centers, LLP, Irving, Texas
  - Texas Oncology San Antonio Medical Center, San Antonio, Texas
  - Texas Oncology, P.A., The Woodlands, Texas
  - Texas Oncology- Northeast Texas, Tyler, Texas
  - Huntsman Cancer Institute; Oncology, Salt Lake City, Utah
  - Dixie Medical Center, St. George, Utah
  - University of Virginia, Charlottesville, Virginia
  - Virginia Cancer Specialists, PC, Fairfax, Virginia
  - Virginia Oncology Associates, Norfolk, Virginia
  - Henrico Doctors' Hospital - Forest, Richmond, Virginia
  - Shenandoah Oncology Associates, Winchester, Virginia
  - University of Washington Seattle Cancer Care Alliance, Seattle, Washington
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - DN Greenwald Center, Mukwonago, Wisconsin
  - Aspirus Regional Cancer Center, Wausau, Wisconsin
- Australia (3):
  - The Royal North Shore Hospital; Northern Sydney Cancer Centre, St Leonards, New South Wales
  - Cabrini Hospital; Cabrini Foundation, Malvern, Victoria
  - Peter MacCallum Cancer Center, North Melbourne, Victoria
- Austria (4):
  - Krankenhaus Der Barmherzigen Brüder Graz; Gynäkologie, Graz
  - Tiroler Landeskrankenanstalten Ges.M.B.H.; Abt. Für Gynäkologie, Innsbruck
  - Landeskrankenhaus Salzburg; Gynäkologie Und Onkologie, Salzburg
  - Medizinische Universität Wien; Univ.Klinik für Frauenheilkunde - Klinik für Gynäkologie, Vienna
- Belgium (4):
  - AZ Maria Middelares, Ghent
  - UZ Gent, Ghent
  - UZ Leuven Gasthuisberg, Leuven
  - Sint Augustinus Wilrijk, Wilrijk
- Brazil (2):
  - Instituto Nacional de Cancer - INCa; Oncologia, Rio de Janeiro, Rio de Janeiro
  - Clinica de Pesquisa e Centro de Estudos em Oncologia Ginecologica e Mamaria Ltda, São Paulo, São Paulo
- China (14):
  - Peking Union Medical College Hospital, Beijing
  - Beijing Cancer Hospital, Beijing
  - West China Second University Hospital, Chengdu
  - Chongqing Cancer Hospital, Chongqing
  - Sun Yet-sen University Cancer Center, Guangzhou
  - Women's hospital school of medicine Zhejiang University, Hangzhou
  - Harbin Medical University Cancer Hospital, Harbin
  - Zhongda Hospital Affiliated to Southeast University, Nanjing
  - Jiangsu Province Hospital (the First Affiliated Hospital With Nanjing Medical University), Nanjing
  - Guangxi Cancer Hospital of Guangxi Medical University, Nanning
  - Fudan University Shanghai Cancer Center, Shanghai
  - Tianjin Central Hospital of Gynecology Obstetrics., Tianjin
  - Zhejiang Cancer Hospital, Zhejiang
  - Henan Cancer Hospital, Zhengzhou
- Czechia (4):
  - Fakultni nemocnice Olomouc; Onkologicka klinika, Olomouc
  - University Hospital Ostrava; Fakultní nemocnice, Ostrava-Poruba
  - Gynekologicko-porodnicka klinika, Prague
  - Onkologicka klinika UK 2.LF a FN v Motole, Prague
- Rigshospitalet; Onkologisk Klinik, København Ø, Denmark
- Finland (3):
  - Kuopio University Hospital, Kuopio
  - Tampereen yliopistollinen sairaala, Tampere
  - Turku Uni Central Hospital; Gynaecology Dept, Turku
- France (8):
  - Clinique Sainte Catherine; Hopital De Semaine, Avignon
  - Ctr Jean Bernard Clin V. Hugo; Service d'Oncologie Méd, Le Mans
  - Centre Léon Bérard; Centre régional; le cancer Rhône-Alpes, Lyon
  - l'Hôpital privé du Confluent SAS, Nantes
  - Hopital Des Diaconesses; Oncologie, Paris
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Centre Rene Huguenin; CONSULT SPECIALISEES, Saint-Cloud
  - Institut Gustave Roussy, Villejuif
- Germany (17):
  - Campus Virchow-Klinikum Charité; Centrum 17; Klinik für Gynäkologie, Berlin
  - Universitätsklinikum Dresden; Klinik für Frauenheilkunde und Geburtshilfe, Dresden
  - Universitätsklinikum Essen; Zentrum Für Frauenheilkunde, Essen
  - Kliniken Essen Mitte Evang. Huyssens Stiftung/Knappschaft GmbH, Essen
  - Universitätsklinikum Freiburg; Frauenklinik, Freiburg im Breisgau
  - Universitätsklinikum Greifswald; Klinik für Frauenheilkunde und Brustzentrum, Greifswald
  - Universitätsklinikum Hamburg-Eppendorf (UKE); Klinik und Poliklinik für Gynäkologie, Hamburg
  - Medizinische Hochschule Hannover, Klinik für Frauenheilkunde und Geburtshilfe, Hanover
  - Universitätsklinikum Heidelberg; Nationales Centrum für Tumorerkrankungen (NCT), Heidelberg
  - Klinikum Konstanz, Frauenklinik, Konstanz
  - Universitätsklinikum Schleswig-Holstein / Campus Lübeck; Klinik für Frauenheilkunde und Geburtshilfe, Lübeck
  - Universitätsmedizin Mainz; Klinik u. Poliklinik f. Geburtshilfe u. Frauenheilkunde, Mainz
  - Klinikum der Universität München; Campus Großhadern; Klinik und Poliklinik für Frauenheilkunde, München
  - Klinikum rechts der Isar der TU München; Klinik und Poliklinik für Frauenheilkunde, München
  - Klinikum Südstadt, Rostock
  - Universitätsklinikum Ulm Am Michelsberg; Frauenklinik, Ulm
  - HELIOS Dr. Horst Schmidt Kliniken Wiesbaden; Klinik für Gynäkologie und gynäkologische Onkologie, Wiesbaden
- Greece (5):
  - Alexandras Hospital; Dept. of Clin. Therapeutics, Athens Uni School of Medicine, Athens
  - Uni Hospital of Ioannina; Oncology Dept., Ioannina
  - Agioi Anargyroi Cancer Hospital; 2Nd Oncology Dept., Kifissia
  - University Hospital of Patras Medical Oncology, Pátrai
  - EUROMEDICA General Clinic of Thessaloniki; Medical Oncology Dept - Oncomedicare, Thessaloniki
- Israel (5):
  - Hillel Yaffe MC; Gynaecology, Hadera
  - Shaare Zedek Medical Center; Oncology Dept, Jerusalem
  - Meir Medical Center; Obstetrics and Gynecology, Kfar Saba
  - Chaim Sheba Medical Center; Obstetrics and Gynecology, Ramat Gan
  - Kaplan Medical Center; Oncology Inst., Rehovot
- Italy (18):
  - Ospedale Antonio Perrino; Oncologia Medica, Brindisi, Apulia
  - Azienda Ospedaliera Universitaria Federico II, Napoli, Campania
  - ISTITUTO NAZIONALE TUMORI IRCCS FONDAZIONE G. PASCALE; Dipartimento Uro-Ginecologico, Napoli, Campania
  - Policlinico S.Orsola-Malpighi; Istituto Oncologia R. Addarii, Bologna, Emilia-Romagna
  - Ospedale Degli Infermi - Faenza; Oncologia Medica, Faenza, Emilia-Romagna
  - IRST Istituto Scientifico Romagnolo Per Lo Studio E Cura Dei Tumori, Sede Meldola; Oncologia Medica, Meldola, Emilia-Romagna
  - Arcispedale Santa Maria Nuova; Oncologia, Reggio Emilia, Emilia-Romagna
  - Policlinico A. Gemelli e C.I.C.; Area Salute della Donna, Rome, Lazio
  - A.O.Spedali Civili; Ostetricia e Ginecologia, Brescia, Lombardy
  - IRCCS S. Raffaele; Ginecologia Oncologica, Milan, Lombardy
  - Istituto Nazionale dei Tumori; Divisione Oncologia Chirurgica e Ginecologica, Milan, Lombardy
  - Irccs Istituto Europeo Di Oncologia (IEO); Oncologia Medica, Milan, Lombardy
  - Asst Grande Ospedale Metropolitano Niguarda; Dipartimento Di Ematologia Ed Oncologia, Milan, Lombardy
  - A.O. San Gerardo; Ginecologia, Monza, Lombardy
  - A. O. Città della Salute e della Scienza; Unità di Oncologia Ginecologica, Turin, Piedmont
  - Ospedale Mauriziano Umberto 1; Ginecologia - Oncologia, Turin, Piedmont
  - Ospedale Silvestrini; Oncologia ed Ematologia, Perugia, Umbria
  - IRCCS Istituto Oncologico Veneto (IOV); Oncologia Medica Seconda, Padua, Veneto
- Japan (22):
  - Nagoya University Hospital, Aichi
  - National Hospital Organization Shikoku Cancer Center, Ehime
  - Ehime University Hospital, Ehime
  - NHO Kyushu Cancer Center, Fukuoka
  - Kyushu University Hospital, Fukuoka
  - Kurume University Hospital, Fukuoka
  - Kure Medical Center, Hiroshima
  - National Hospital Organization Hokkaido Cancer Center, Hokkaido
  - Hyogo Cancer Center, Hyōgo
  - Kagoshima University Hospital, Kagoshima
  - Yokohama City University Hospital, Kanagawa
  - Kyoto University Hospital, Kyoto
  - Mie University Hospital, Mie
  - Tohoku University Hospital, Miyagi
  - Niigata University Medical & Dental Hospital, Niigata
  - Iwate Medical University Hospital, Numakunai
  - Osaka International Cancer Institute, Osaka
  - Shizuoka Cancer Center, Shizuoka
  - The Jikei University Hospital, Tokyo
  - The University of Tokyo Hospital, Tokyo
  - The Cancer Institute Hospital of JFCR, Tokyo
  - Keio University Hospital, Tokyo
- Norway (2):
  - Oslo Universitetssykehus HF; Radiumhospitalet, Oslo
  - St. Olavs Hospital, Trondheim
- Poland (4):
  - Centrum Onkologii Instytut im. M.Sklodowskiej-Curie; Klinika Ginekologii Onkologicznej, Krakow
  - Szpital Kliniczny im. Heliodora ?wi?cickiego UM w Poznaniu; Oddzia? Ginekologii Onkologicznej, Późna
  - Icu Spsk - 2, Szczecin
  - Narodowy Instytut Onkologii im. M.Sklodowskiej-Curie;Klinika Ginekologii Onkologicznej, Warsaw
- Russia (4):
  - Moscow City Oncology Hospital #62, Moscovskaya Oblast, Moscow Oblast
  - Clinical Oncology Dispensary of Ministry of Health of Tatarstan, Kazan'
  - N.N.Burdenko Main Military Clinical Hospital; Oncology Dept, Moscow
  - St. Petersburg Oncology & Gynecology; City Clinical Oncology Dispensary, Saint Petersburg
- South Korea (4):
  - National Cancer Center, Goyang-si
  - Seoul National University Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
- Spain (9):
  - Hospital Universitario Son Espases, Palma de Mallorca, Balearic Islands
  - Corporacio Sanitaria Parc Tauli; Servicio de Oncologia, Sabadell, Barcelona
  - Fundacion Hospital de Alcorcon; Servicio de Oncologia, Alcorcón, Madrid
  - Hospital Universitari Dexeus - Grupo Quironsalud; Servicio de Oncologia Medica, Barcelona
  - Hospital General Universitario Gregorio Marañon; Servicio de Oncologia, Madrid
  - Centro Integral Oncologico Clara Campal; Servicio de Oncología, Madrid
  - Hospital Clinico Universitario Virgen de la Victoria; Servicio de Oncologia, Málaga
  - Hospital Universitario la Fe; Servicio de Oncologia, Valencia
  - Hospital Universitario Miguel Servet; Servicio Oncologia, Zaragoza
- Sweden (2):
  - Uni Hospital Linkoeping; Dept. of Oncology, Linköping
  - Karolinska Hospital; Oncology - Radiumhemmet, Stockholm
- Turkey (Türkiye) (6):
  - Baskent University Adana Dr. Turgut Noyan Practice and Research Hospital; Medical Oncology, Adana
  - Ankara University Medical Faculty; Medikal Onkoloji, Ankara
  - Baskent Universitesi Ankara Hastanesi; T?bbi Onkoloji Bölümü, Ankara
  - Koc University Medical Faculty; Department of Gynecology & Obstetrics, Istanbul
  - Istanbul Uni Istanbul Medical Faculty, Istanbul
  - Istanbul University Cerrahpasa Medical Faculty; Obstetrics and Gynecology, Istanbul

REFERENCES:
- [Derived] Pignata S, Bookman M, Sehouli J, Miller A, Penson RT, Taskiran C, Anderson C, Hietanen S, Myers T, Madry R, Willmott L, Lortholary A, Thomes-Pepin J, Aghajanian C, McCourt C, Stuckey A, Wu X, Nishio S, Copeland LJ, He Y, Molinero L, Patel S, Lin YG, Khor VK, Moore KN. Overall survival and patient-reported outcome results from the placebo-controlled randomized phase III IMagyn050/GOG 3015/ENGOT-OV39 trial of atezolizumab for newly diagnosed stage III/IV ovarian cancer. Gynecol Oncol. 2023 Oct;177:20-31. doi: 10.1016/j.ygyno.2023.06.018. Epub 2023 Aug 23. PMID 37625235
- [Derived] Landen CN, Molinero L, Hamidi H, Sehouli J, Miller A, Moore KN, Taskiran C, Bookman M, Lindemann K, Anderson C, Berger R, Myers T, Beiner M, Reid T, Van Nieuwenhuysen E, Green A, Okamoto A, Aghajanian C, Thaker PH, Blank SV, Khor VK, Chang CW, Lin YG, Pignata S. Influence of Genomic Landscape on Cancer Immunotherapy for Newly Diagnosed Ovarian Cancer: Biomarker Analyses from the IMagyn050 Randomized Clinical Trial. Clin Cancer Res. 2023 May 1;29(9):1698-1707. doi: 10.1158/1078-0432.CCR-22-2032. PMID 36595569
- [Derived] Moore KN, Bookman M, Sehouli J, Miller A, Anderson C, Scambia G, Myers T, Taskiran C, Robison K, Maenpaa J, Willmott L, Colombo N, Thomes-Pepin J, Liontos M, Gold MA, Garcia Y, Sharma SK, Darus CJ, Aghajanian C, Okamoto A, Wu X, Safin R, Wu F, Molinero L, Maiya V, Khor VK, Lin YG, Pignata S. Atezolizumab, Bevacizumab, and Chemotherapy for Newly Diagnosed Stage III or IV Ovarian Cancer: Placebo-Controlled Randomized Phase III Trial (IMagyn050/GOG 3015/ENGOT-OV39). J Clin Oncol. 2021 Jun 10;39(17):1842-1855. doi: 10.1200/JCO.21.00306. Epub 2021 Apr 23. PMID 33891472
- [Derived] Moore KN, Pignata S; IMagyn050 Steering Committee. Trials in progress: IMagyn050/GOG 3015/ENGOT-OV39. A Phase III, multicenter, randomized study of atezolizumab versus placebo administered in combination with paclitaxel, carboplatin, and bevacizumab to patients with newly-diagnosed stage III or stage IV ovarian, fallopian tube, or primary peritoneal cancer. Int J Gynecol Cancer. 2019 Feb 4;29(2):430-433. doi: 10.1136/ijgc-2018-000071. PMID 30630885

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study is considered "Completed" because all pre-planned study activities and analyses have been performed.
Groups:
- Placebo With Paclitaxel, Carboplatin and Bevacizumab: Participants in the primary tumor-reductive surgery group received paclitaxel, carboplatin, atezolizumab placebo IV infusion on Day 1 of each 21-day cycle for a total of 6 cycles, and bevacizumab IV infusion starting with Cycle 2 for a total of 5 cycles, followed by maintenance therapy bevacizumab with atezolizumab placebo for a total of 22 cycles of atezolizumab placebo and 21 cycles of bevacizumab. Participants in the neoadjuvant therapy group received paclitaxel, carboplatin and placebo for 6 cycles and bevacizumab for 4 cycles. Interval surgery will occur between cycles 3 and 4. Each cycle is 21 days long. After 6 cycles, participants started maintenance therapy of bevacizumab and placebo for additional 16 cycles.
- Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab: Participants in the primary tumor-reductive surgery group received paclitaxel, carboplatin, atezolizumab intravenous (IV) infusion on Day 1 of each 21-day cycle for a total of 6 cycles, and bevacizumab IV infusion starting with Cycle 2 for a total of 5 cycles, followed by maintenance therapy bevacizumab with atezolizumab for a total of 22 cycles of atezolizumab and 21 cycles of bevacizumab. Participants in the neoadjuvant therapy group received paclitaxel, carboplatin and atezolizumab for 6 cycles and bevacizumab for 4 cycles. Interval surgery will occur between cycles 3 and 4. Each cycle is 21 days long. After 6 cycles, participants started maintenance therapy of bevacizumab and atezolizumab for additional 16 cycles.
Period: Overall Study
Arm/Group | Placebo With Paclitaxel, Carboplatin and Bevacizumab | Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab
Started | 650 | 651
Completed | 0 | 0
Not Completed | 650 | 651
Not completed — Death | 289 | 272
Not completed — Lost to Follow-up | 9 | 10
Not completed — Protocol Deviation | 1 | 4
Not completed — Withdrawal by Subject | 45 | 51
Not completed — Study Terminated By Sponsor | 305 | 311
Not completed — Physician Decision | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo With Paclitaxel, Carboplatin and Bevacizumab | Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab | Total
Number analyzed (Participants) | 650 | 651 | 1301
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.3 (10.7) | 58.9 (10.5) | 59.1 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 650 | 651 | 1301
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 38 | 39 | 77
  Not Hispanic or Latino | 598 | 589 | 1187
  Unknown or Not Reported | 14 | 23 | 37
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 6 | 5 | 11
  Asian | 155 | 150 | 305
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 2
  Black or African American | 13 | 8 | 21
  White | 461 | 464 | 925
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 15 | 22 | 37

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS) Assessed by Investigator as Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) - Intent-to-Treat (ITT) Population
Description: Investigator-assessed PFS is defined as the time from randomization to the occurrence of disease progression, as determined by the investigator from tumor assessments per RECIST v1.1, or death from any cause during the study, whichever occurs first.
Time Frame: From randomization until disease progression or death from any cause (up to approximately 55 months)
Population: Intent-to-Treat (ITT) population is defined as all randomized patients, whether or not the assigned study treatment was received.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Placebo With Paclitaxel, Carboplatin and Bevacizumab | Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab
Number analyzed (Participants) | 650 | 651
Months | 18.37 [17.22 to 19.75] | 19.48 [18.14 to 20.76]
Statistical Analysis 1: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Test type: Superiority; p = 0.2785, Log Rank; Hazard Ratio (HR) = 0.92, 95% CI 2-sided [0.79 to 1.07]

2. Primary Outcome: PFS Assessed by Investigator as Per RECIST v1.1 - Programmed Death-Ligand 1 (PD-L1)-Positive Subpopulation
Description: as for outcome 1
Time Frame: From randomization until disease progression or death from any cause (up to approximately 55 months)
Population: PD-L1-positive subpopulation is defined as patients in the ITT population whose PD-L1 status was IC1/2/3 at the time of randomization.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Placebo With Paclitaxel, Carboplatin and Bevacizumab | Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab
Number analyzed (Participants) | 393 | 391
Months | 18.50 [16.62 to 21.36] | 20.83 [19.06 to 24.21]
Statistical Analysis 1: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Test type: Superiority — Stratified Analysis; p = 0.0376, Log Rank; Hazard Ratio (HR) = 0.80, 95% CI 2-sided [0.65 to 0.99]

3. Primary Outcome: Overall Survival - ITT Population
Description: Overall Survival (OS) is defined as the time from randomization to death from any cause.
Time Frame: From randomization up to death from any cause (up to approximately 59 months)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Placebo With Paclitaxel, Carboplatin and Bevacizumab | Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab
Number analyzed (Participants) | 650 | 651
Months | 46.59 [45.31 to 49.74] | 50.53 [46.26 to NA] — The upper limit of 95% CI was not estimable by Brookmeyer and Crowley method due to insufficient observed events.
Statistical Analysis 1: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Stratified by: stage and/or surgical status (Stage III vs. Stage IV), ECOG performance status (0 vs. 1 or 2), tumor PD-L1 status (IC0 vs. IC1/2/3), and treatment strategy (adjuvant vs. neoadjuvant); Test type: Superiority; p = 0.3432, Log Rank; Hazard Ratio (HR) = 0.92, 95% CI 2-sided [0.78 to 1.09]

4. Primary Outcome: Overall Survival - PD-L1-Positive Subpopulation
Description: Overall Survival (OS) is defined as the time from randomization to death from any cause.
Time Frame: From randomization up to death from any cause (up to approximately 59 months)
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Placebo With Paclitaxel, Carboplatin and Bevacizumab | Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab
Number analyzed (Participants) | 393 | 391
Months | 49.15 [45.54 to NA] — The upper limit of 95% CI was not estimable by Brookmeyer and Crowley method due to insufficient observed events. | NA [NA to NA] — 67.3% of the participants were censored and the median was not reached.
Statistical Analysis 1: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Stratified by: stage and/or surgical status (Stage III vs. Stage IV), ECOG performance status (0 vs. 1 or 2) and treatment strategy (adjuvant vs. neoadjuvant); Test type: Superiority — Stratified Analysis; p = 0.1316, Log Rank; Hazard Ratio (HR) = 0.83, 95% CI 2-sided [0.66 to 1.06]

5. Secondary Outcome: Percentage of Participants With Objective Response (OR) Assessed by Investigator as Per RECIST v1.1 - Primary Tumor-Reductive Surgery Group in ITT Population
Description: OR is defined as either a CR or PR as determined by the investigator with the use of RECIST v1.1 for patients with measurable residual disease after primary surgery.
Time Frame: From randomization until disease progression or death from any cause (up to approximately 55 months)
Population: Objective Response Rate (ORR) - evaluable population is defined as primary surgery patients in the ITT population with measurable disease at baseline.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo With Paclitaxel, Carboplatin and Bevacizumab | Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab
Number analyzed (Participants) | 650 | 651
Percentage of participants | 88.7 | 92.8

6. Secondary Outcome: Percentage of Participants With Objective Response (OR) Assessed by Investigator as Per RECIST v1.1 - Primary Tumor-Reductive Surgery Group in PD-L1-Positive Population
Description: as for outcome 5
Time Frame: From randomization until disease progression or death from any cause (up to approximately 55 months)
Population: Objective Response Rate (ORR) - evaluable population is defined as primary surgery patients in the PD-L1-Positive subpopulation with measurable disease at baseline.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo With Paclitaxel, Carboplatin and Bevacizumab | Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab
Number analyzed (Participants) | 393 | 391
Percentage of participants | 89.9 | 92.3

7. Secondary Outcome: Duration of Response Assessed by Investigator as Per RECIST v1.1 - Primary Tumor-Reductive Surgery (Having Residual Measurable Disease) Group in ITT Population
Description: DOR is defined as the time interval from first occurrence of a CR or PR to the time of disease progression, as determined by the investigator with the use of RECIST v1.1, or death from any cause, whichever comes first for patients with measurable residual disease after primary surgery.
Time Frame: From the date of first occurrence of a confirmed complete or partial response until disease progression or death from any cause (up to approximately 55 months)
Population: Duration of Objective Response (DOR) - evaluable population is defined as patients with an objective response. The ITT population is defined as all randomized patients, whether or not the assigned study treatment was received.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Placebo With Paclitaxel, Carboplatin and Bevacizumab | Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab
Number analyzed (Participants) | 650 | 651
Months | 14.06 [13.01 to 16.62] | 16.59 [14.52 to 19.09]

8. Secondary Outcome: Duration of Response Assessed by Investigator as Per RECIST v1.1 - Primary Tumor-Reductive Surgery (Having Residual Measurable Disease) Group in PD-L1-Positive Population
Description: as for outcome 7
Time Frame: as for outcome 7
Population: Duration of Objective Response (DOR) - evaluable population is defined as patients with an objective response. The PD-L1-positive subpopulation (defined as patients in the ITT population whose PD-L1 status is IC1/2/3 at the time of randomization) who underwent primary tumor-reductive surgery.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Placebo With Paclitaxel, Carboplatin and Bevacizumab | Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab
Number analyzed (Participants) | 142 | 156
Months | 13.44 [12.71 to 19.29] | 17.71 [15.01 to 19.61]

9. Secondary Outcome: Percentage of Participants Who Achieve a Clinically-Meaningful Improvement in Patient-Reported Abdominal Pain and Bloating - Neoadjuvant Group
Description: Clinically-meaningful improvement defined as a >=10-point decrease from the baseline score in patient-reported abdominal pain or bloating will be assessed using European Organisation for Research and Treatment of Cancer Quality-of-Life Questionnaires Ovarian Cancer Module 28 (EORTC QLQ-OV28) Abdominal/Gastrointestinal Symptom Scale (Items 31 and 31).
Time Frame: From randomization to the end of treatment/discontinuation (up to approximately 66 weeks), and during follow-up period (up to approximately 55 months). Cycle length=21 days.
Population: Neoadjuvant Group. PRO-evaluable population is defined as patients in the ITT population with a baseline and >=1 post-baseline PRO assessment. The ITT population is defined as all randomized patients, whether or not the assigned study treatment was received.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo With Paclitaxel, Carboplatin and Bevacizumab | Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab
Number analyzed (Participants) | 157 | 152
Percentage of participants
  Abdominal Pain, Presurgical/Surgery: number analyzed (Participants) | 142 | 136
  Abdominal Pain, Presurgical/Surgery | 54.2 | 50.7
  Abdominal Pain, Cycle 4 Day 1: number analyzed (Participants) | 140 | 133
  Abdominal Pain, Cycle 4 Day 1 | 36.4 | 32.3
  Abdominal Pain, Cycle 6 Day 1: number analyzed (Participants) | 131 | 133
  Abdominal Pain, Cycle 6 Day 1 | 55.0 | 48.1
  Abdominal Pain, Cycle 8 Day 1: number analyzed (Participants) | 129 | 122
  Abdominal Pain, Cycle 8 Day 1 | 64.3 | 54.1
  Abdominal Pain, Cycle 12 Day 1: number analyzed (Participants) | 111 | 101
  Abdominal Pain, Cycle 12 Day 1 | 63.1 | 57.4
  Abdominal Pain, Cycle 16 Day 1: number analyzed (Participants) | 96 | 88
  Abdominal Pain, Cycle 16 Day 1 | 63.5 | 58.0
  Abdominal Pain, Cycle 20 Day 1: number analyzed (Participants) | 83 | 62
  Abdominal Pain, Cycle 20 Day 1 | 68.7 | 48.4
  Abdominal Pain, Completion of Treatment/Early Termination Visit: number analyzed (Participants) | 143 | 130
  Abdominal Pain, Completion of Treatment/Early Termination Visit | 51.0 | 51.5
  Abdominal Pain, Post-Treatment Follow Up 3 Months: number analyzed (Participants) | 96 | 96
  Abdominal Pain, Post-Treatment Follow Up 3 Months | 58.3 | 51.0
  Abdominal Pain, Post-Treatment Follow Up 6 Months: number analyzed (Participants) | 75 | 74
  Abdominal Pain, Post-Treatment Follow Up 6 Months | 61.3 | 51.4
  Abdominal Pain, Post-Treatment Follow Up 9 Months: number analyzed (Participants) | 43 | 38
  Abdominal Pain, Post-Treatment Follow Up 9 Months | 60.5 | 50.0
  Abdominal Pain, Post-Treatment Follow Up 12 Months: number analyzed (Participants) | 17 | 24
  Abdominal Pain, Post-Treatment Follow Up 12 Months | 70.6 | 58.3
  Abdominal Pain, Post-Treatment Follow Up 18 Months: number analyzed (Participants) | 6 | 4
  Abdominal Pain, Post-Treatment Follow Up 18 Months | 100 | 50.0
  Abdominal Pain, Post-Treatment Follow Up 24 Months: number analyzed (Participants) | 1 | 2
  Abdominal Pain, Post-Treatment Follow Up 24 Months | 100 | 100
  Bloating, Presurgical/Surgery: number analyzed (Participants) | 142 | 137
  Bloating, Presurgical/Surgery | 62.7 | 54.0
  Bloating, Cycle 4 Day 1: number analyzed (Participants) | 140 | 132
  Bloating, Cycle 4 Day 1 | 65.0 | 59.8
  Bloating, Cycle 6 Day 1: number analyzed (Participants) | 131 | 133
  Bloating, Cycle 6 Day 1 | 71.0 | 66.9
  Bloating, Cycle 8 Day 1: number analyzed (Participants) | 128 | 123
  Bloating, Cycle 8 Day 1 | 71.9 | 63.4
  Bloating, Cycle 12 Day 1: number analyzed (Participants) | 111 | 101
  Bloating, Cycle 12 Day 1 | 68.5 | 63.4
  Bloating, Cycle 16 Day 1: number analyzed (Participants) | 96 | 88
  Bloating, Cycle 16 Day 1 | 66.7 | 64.8
  Bloating, Cycle 20 Day 1: number analyzed (Participants) | 83 | 62
  Bloating, Cycle 20 Day 1 | 66.3 | 56.5
  Bloating, Completion of Treatment/ Early Termination Visit: number analyzed (Participants) | 145 | 130
  Bloating, Completion of Treatment/ Early Termination Visit | 62.1 | 58.5
  Bloating, Post-Treatment Follow Up 3 Months: number analyzed (Participants) | 96 | 96
  Bloating, Post-Treatment Follow Up 3 Months | 57.3 | 53.1
  Bloating, Post-Treatment Follow Up 6 Months: number analyzed (Participants) | 76 | 74
  Bloating, Post-Treatment Follow Up 6 Months | 59.2 | 62.2
  Bloating, Post-Treatment Follow Up 9 Months: number analyzed (Participants) | 43 | 38
  Bloating, Post-Treatment Follow Up 9 Months | 67.4 | 63.2
  Bloating, Post-Treatment Follow Up 12 Months: number analyzed (Participants) | 17 | 24
  Bloating, Post-Treatment Follow Up 12 Months | 47.1 | 62.5
  Bloating, Post-Treatment Follow Up 18 Months: number analyzed (Participants) | 6 | 4
  Bloating, Post-Treatment Follow Up 18 Months | 66.7 | 50.0
  Bloating, Post-Treatment Follow Up 24 Months: number analyzed (Participants) | 1 | 2
  Bloating, Post-Treatment Follow Up 24 Months | 0 | 100

10. Secondary Outcome: Percentage of Participants Who Achieve a Clinically-Meaningful Improvement in Patient-Reported Function and Health Related Quality of Life (HRQoL) - Neoadjuvant Group
Description: Clinically-meaningful improvement in patient-reported function and HRQoL during the treatment period, defined as a >=10-point increase from the baseline score on each of the functional (social, emotional, physical, role) and GHS/QoLscales of the European Organisation for Research and Treatment of Cancer Quality-of-Life Questionnaires Core 30 (EORTC QLQ-C30).
Time Frame: as for outcome 9
Population: PRO-evaluable population is defined as patients in the ITT population with a baseline and >=1 post-baseline PRO assessment.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo With Paclitaxel, Carboplatin and Bevacizumab | Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab
Number analyzed (Participants) | 157 | 152
Percentage of participants
  Physical Functioning, Presurgical/Surgery: number analyzed (Participants) | 142 | 137
  Physical Functioning, Presurgical/Surgery | 35.9 | 33.6
  Physical Functioning, Cycle 4 Day 1: number analyzed (Participants) | 141 | 133
  Physical Functioning, Cycle 4 Day 1 | 28.4 | 18.0
  Physical Functioning, Cycle 6 Day 1: number analyzed (Participants) | 132 | 133
  Physical Functioning, Cycle 6 Day 1 | 35.6 | 25.6
  Physical Functioning, Cycle 8 Day 1: number analyzed (Participants) | 129 | 123
  Physical Functioning, Cycle 8 Day 1 | 37.2 | 36.6
  Physical Functioning, Cycle 12 Day 1: number analyzed (Participants) | 111 | 102
  Physical Functioning, Cycle 12 Day 1 | 45.9 | 43.1
  Physical Functioning, Cycle 16 Day 1: number analyzed (Participants) | 96 | 88
  Physical Functioning, Cycle 16 Day 1 | 42.7 | 42.0
  Physical Functioning, Cycle 20 Day 1: number analyzed (Participants) | 83 | 63
  Physical Functioning, Cycle 20 Day 1 | 41.0 | 31.7
  Physical Functioning, Completion of Treatment/Early Termination Visit: number analyzed (Participants) | 144 | 131
  Physical Functioning, Completion of Treatment/Early Termination Visit | 38.9 | 34.4
  Physical Functioning, Post-Treatment Follow Up 3 Months: number analyzed (Participants) | 97 | 97
  Physical Functioning, Post-Treatment Follow Up 3 Months | 37.1 | 39.2
  Physical Functioning, Post-Treatment Follow Up 6 Months: number analyzed (Participants) | 76 | 74
  Physical Functioning, Post-Treatment Follow Up 6 Months | 40.8 | 39.2
  Physical Functioning, Post-Treatment Follow Up 9 Months: number analyzed (Participants) | 43 | 38
  Physical Functioning, Post-Treatment Follow Up 9 Months | 32.6 | 50.0
  Physical Functioning, Post-Treatment Follow Up 12 Months: number analyzed (Participants) | 17 | 24
  Physical Functioning, Post-Treatment Follow Up 12 Months | 23.5 | 37.5
  Physical Functioning, Post-Treatment Follow Up 18 Months: number analyzed (Participants) | 6 | 4
  Physical Functioning, Post-Treatment Follow Up 18 Months | 33.3 | 50.0
  Physical Functioning, Post-Treatment Follow Up 24 Months: number analyzed (Participants) | 1 | 2
  Physical Functioning, Post-Treatment Follow Up 24 Months | 100 | 50.0
  Role Functioning, Presurgical/Surgery: number analyzed (Participants) | 142 | 137
  Role Functioning, Presurgical/Surgery | 48.6 | 40.9
  Role Functioning, Cycle 4 Day 1: number analyzed (Participants) | 141 | 133
  Role Functioning, Cycle 4 Day 1 | 38.3 | 22.6
  Role Functioning, Cycle 6 Day 1: number analyzed (Participants) | 133 | 134
  Role Functioning, Cycle 6 Day 1 | 45.9 | 33.6
  Role Functioning, Cycle 8 Day 1: number analyzed (Participants) | 129 | 123
  Role Functioning, Cycle 8 Day 1 | 50.4 | 39.8
  Role Functioning, Cycle 12 Day 1: number analyzed (Participants) | 111 | 102
  Role Functioning, Cycle 12 Day 1 | 55.9 | 47.1
  Role Functioning, Cycle 16 Day 1: number analyzed (Participants) | 96 | 88
  Role Functioning, Cycle 16 Day 1 | 53.1 | 46.6
  Role Functioning, Cycle 20 Day 1: number analyzed (Participants) | 83 | 63
  Role Functioning, Cycle 20 Day 1 | 56.6 | 52.4
  Role Functioning, Completion of Treatment/ Early Termination Visit: number analyzed (Participants) | 145 | 131
  Role Functioning, Completion of Treatment/ Early Termination Visit | 46.9 | 39.7
  Role Functioning, Post-Treatment Follow Up 3 Months: number analyzed (Participants) | 97 | 97
  Role Functioning, Post-Treatment Follow Up 3 Months | 49.5 | 40.2
  Role Functioning, Post-Treatment Follow Up 6 Months: number analyzed (Participants) | 76 | 74
  Role Functioning, Post-Treatment Follow Up 6 Months | 51.3 | 48.6
  Role Functioning, Post-Treatment Follow Up 9 Months: number analyzed (Participants) | 43 | 38
  Role Functioning, Post-Treatment Follow Up 9 Months | 53.5 | 52.6
  Role Functioning, Post-Treatment Follow Up 12 Months: number analyzed (Participants) | 17 | 24
  Role Functioning, Post-Treatment Follow Up 12 Months | 23.5 | 54.2
  Role Functioning, Post-Treatment Follow Up 18 Months: number analyzed (Participants) | 6 | 4
  Role Functioning, Post-Treatment Follow Up 18 Months | 50.0 | 50.0
  Role Functioning, Post-Treatment Follow Up 24 Months: number analyzed (Participants) | 1 | 2
  Role Functioning, Post-Treatment Follow Up 24 Months | 0 | 50.0
  Social Functioning, Presurgical/Surgery: number analyzed (Participants) | 142 | 137
  Social Functioning, Presurgical/Surgery | 32.4 | 33.6
  Social Functioning, Cycle 4 Day 1: number analyzed (Participants) | 141 | 133
  Social Functioning, Cycle 4 Day 1 | 31.2 | 25.6
  Social Functioning, Cycle 6 Day 1: number analyzed (Participants) | 133 | 132
  Social Functioning, Cycle 6 Day 1 | 36.8 | 33.3
  Social Functioning, Cycle 8 Day 1: number analyzed (Participants) | 129 | 122
  Social Functioning, Cycle 8 Day 1 | 40.3 | 39.3
  Social Functioning, Cycle 12 Day 1: number analyzed (Participants) | 111 | 101
  Social Functioning, Cycle 12 Day 1 | 39.6 | 44.6
  Social Functioning, Cycle 16 Day 1: number analyzed (Participants) | 95 | 88
  Social Functioning, Cycle 16 Day 1 | 40.0 | 44.3
  Social Functioning, Cycle 20 Day 1: number analyzed (Participants) | 83 | 62
  Social Functioning, Cycle 20 Day 1 | 45.8 | 43.5
  Social Functioning, Completion of Treatment/Early Termination: number analyzed (Participants) | 144 | 130
  Social Functioning, Completion of Treatment/Early Termination | 40.3 | 41.5
  Social Functioning, Post-Treatment Follow Up 3 Months: number analyzed (Participants) | 96 | 96
  Social Functioning, Post-Treatment Follow Up 3 Months | 42.7 | 44.8
  Social Functioning, Post-Treatment Follow Up 6 Months: number analyzed (Participants) | 76 | 74
  Social Functioning, Post-Treatment Follow Up 6 Months | 46.1 | 35.1
  Social Functioning, Post-Treatment Follow Up 9 Months: number analyzed (Participants) | 43 | 38
  Social Functioning, Post-Treatment Follow Up 9 Months | 46.5 | 47.4
  Social Functioning, Post-Treatment Follow Up 12 Months: number analyzed (Participants) | 17 | 24
  Social Functioning, Post-Treatment Follow Up 12 Months | 29.4 | 54.2
  Social Functioning, Post-Treatment Follow Up 18 Months: number analyzed (Participants) | 6 | 4
  Social Functioning, Post-Treatment Follow Up 18 Months | 66.7 | 75.0
  Social Functioning, Post-Treatment Follow Up 24 Months: number analyzed (Participants) | 1 | 2
  Social Functioning, Post-Treatment Follow Up 24 Months | 0 | 50.0
  Emotional Functioning, Presurgical/Surgery: number analyzed (Participants) | 142 | 137
  Emotional Functioning, Presurgical/Surgery | 31.7 | 30.7
  Emotional Functioning, Cycle 4 Day 1: number analyzed (Participants) | 141 | 132
  Emotional Functioning, Cycle 4 Day 1 | 31.2 | 35.6
  Emotional Functioning, Cycle 6 Day 1: number analyzed (Participants) | 133 | 131
  Emotional Functioning, Cycle 6 Day 1 | 42.1 | 38.2
  Emotional Functioning, Cycle 8 Day 1: number analyzed (Participants) | 129 | 123
  Emotional Functioning, Cycle 8 Day 1 | 39.5 | 44.7
  Emotional Functioning, Cycle 12 Day 1: number analyzed (Participants) | 111 | 101
  Emotional Functioning, Cycle 12 Day 1 | 41.4 | 41.6
  Emotional Functioning, Cycle 16 Day 1: number analyzed (Participants) | 96 | 88
  Emotional Functioning, Cycle 16 Day 1 | 44.8 | 42.0
  Emotional Functioning, Cycle 20 Day 1: number analyzed (Participants) | 83 | 62
  Emotional Functioning, Cycle 20 Day 1 | 44.6 | 32.3
  Emotional Functioning, Completion of Treatment/Early Termination Visit: number analyzed (Participants) | 145 | 130
  Emotional Functioning, Completion of Treatment/Early Termination Visit | 33.8 | 33.8
  Emotional Functioning, Post-Treatment Follow Up 3 months: number analyzed (Participants) | 96 | 96
  Emotional Functioning, Post-Treatment Follow Up 3 months | 35.4 | 33.3
  Emotional Functioning, Post-Treatment Follow Up 6 months: number analyzed (Participants) | 76 | 74
  Emotional Functioning, Post-Treatment Follow Up 6 months | 30.3 | 33.8
  Emotional Functioning, Post-Treatment Follow Up 9 months: number analyzed (Participants) | 43 | 38
  Emotional Functioning, Post-Treatment Follow Up 9 months | 39.5 | 34.2
  Emotional Functioning, Post-Treatment Follow Up 12 months: number analyzed (Participants) | 17 | 24
  Emotional Functioning, Post-Treatment Follow Up 12 months | 29.4 | 29.2
  Emotional Functioning, Post-Treatment Follow Up 18 months: number analyzed (Participants) | 6 | 4
  Emotional Functioning, Post-Treatment Follow Up 18 months | 16.7 | 50.0
  Emotional Functioning, Post-Treatment Follow Up 24 months: number analyzed (Participants) | 1 | 2
  Emotional Functioning, Post-Treatment Follow Up 24 months | 0 | 50.0
  GHS/HRQoL, PresurgicalSurgery: number analyzed (Participants) | 142 | 137
  GHS/HRQoL, PresurgicalSurgery | 44.4 | 46.7
  GHS/HRQoL, Cycle 4 Day 1: number analyzed (Participants) | 141 | 132
  GHS/HRQoL, Cycle 4 Day 1 | 43.3 | 37.1
  GHS/HRQoL, Cycle 6 Day 1: number analyzed (Participants) | 133 | 132
  GHS/HRQoL, Cycle 6 Day 1 | 51.1 | 47.7
  GHS/HRQoL, Cycle 8 Day 1: number analyzed (Participants) | 129 | 122
  GHS/HRQoL, Cycle 8 Day 1 | 55.0 | 59.0
  GHS/HRQoL, Cycle 12 Day 1: number analyzed (Participants) | 111 | 101
  GHS/HRQoL, Cycle 12 Day 1 | 60.4 | 61.4
  GHS/HRQoL, Cycle 16 Day 1: number analyzed (Participants) | 96 | 88
  GHS/HRQoL, Cycle 16 Day 1 | 53.1 | 58.0
  GHS/HRQoL, Cycle 20 Day 1: number analyzed (Participants) | 83 | 62
  GHS/HRQoL, Cycle 20 Day 1 | 59.0 | 61.3
  GHS/HRQoL, Completion of Treatment/ Early Termination Visit: number analyzed (Participants) | 145 | 130
  GHS/HRQoL, Completion of Treatment/ Early Termination Visit | 46.9 | 53.1
  GHS/HRQoL, Post-Treatment Follow Up 3 Months: number analyzed (Participants) | 95 | 96
  GHS/HRQoL, Post-Treatment Follow Up 3 Months | 53.7 | 53.1
  GHS/HRQoL, Post-Treatment Follow Up 6 Months: number analyzed (Participants) | 76 | 74
  GHS/HRQoL, Post-Treatment Follow Up 6 Months | 48.7 | 41.9
  GHS/HRQoL, Post-Treatment Follow Up 9 Months: number analyzed (Participants) | 43 | 38
  GHS/HRQoL, Post-Treatment Follow Up 9 Months | 39.5 | 50.0
  GHS/HRQoL, Post-Treatment Follow Up 12 Months: number analyzed (Participants) | 17 | 24
  GHS/HRQoL, Post-Treatment Follow Up 12 Months | 17.6 | 41.7
  GHS/HRQoL, Post-Treatment Follow Up 18 Months: number analyzed (Participants) | 6 | 4
  GHS/HRQoL, Post-Treatment Follow Up 18 Months | 16.7 | 50.0
  GHS/HRQoL, Post-Treatment Follow Up 24 Months: number analyzed (Participants) | 1 | 2
  GHS/HRQoL, Post-Treatment Follow Up 24 Months | 0 | 50.0
Statistical Analysis 1: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Emotional Functioning, Presurgical/Surgery; Test type: Superiority — Stratified Analysis; p = 0.9096, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.97, 95% CI 2-sided [0.58 to 1.62]
Statistical Analysis 2: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Emotional functioning, Cycle 4 Day 1; Test type: Superiority — Stratified Analysis; p = 0.4662, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.21, 95% CI 2-sided [0.73 to 2.01]
Statistical Analysis 3: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Emotional functioning, Cycle 6 Day 1; Test type: Superiority — Stratified Analysis; p = 0.5237, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.85, 95% CI 2-sided [0.51 to 1.40]
Statistical Analysis 4: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Emotional functioning, Cycle 8 Day 1; Test type: Superiority — Stratified Analysis; p = 0.3826, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.25, 95% CI 2-sided [0.76 to 2.07]
Statistical Analysis 5: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Emotional Functioning, Cycle 12 Day 1; Test type: Superiority — Stratified Analysis; p = 0.9893, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.00, 95% CI 2-sided [0.56 to 1.76]
Statistical Analysis 6: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Emotional Functioning, Cycle 16 Day 1; Test type: Superiority — Stratified Analysis; p = 0.6892, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.89, 95% CI 2-sided [0.49 to 1.61]
Statistical Analysis 7: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Emotional Functioning, Cycle 20 Day 1; Test type: Superiority — Stratified Analysis; p = 0.1324, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.59, 95% CI 2-sided [0.30 to 1.17]
Statistical Analysis 8: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Emotional Functioning, Completion of Treatment/Early Termination Visit; Test type: Superiority — Stratified Analysis; p = 0.9176, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.03, 95% CI 2-sided [0.62 to 1.70]
Statistical Analysis 9: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Emotional Functioning, Post-Treatment Follow Up 3 Months; Test type: Superiority — Stratified Analysis; p = 0.7861, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.92, 95% CI 2-sided [0.50 to 1.68]
Statistical Analysis 10: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Emotional Functioning, Post-Treatment Follow Up 6 Months; Test type: Superiority — Stratified Analysis; p = 0.4539, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.31, 95% CI 2-sided [0.65 to 2.65]
Statistical Analysis 11: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Emotional Functioning, Post-Treatment Follow Up 9 Months; Test type: Superiority — Stratified Analysis; p = 0.4849, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.71, 95% CI 2-sided [0.27 to 1.86]
Statistical Analysis 12: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Emotional Functioning, Post-Treatment Follow Up 12 Months; Test type: Superiority — Stratified Analysis; p = 0.7470, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.79, 95% CI 2-sided [0.19 to 3.34]
Statistical Analysis 13: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Emotional Functioning, Post-Treatment Follow Up 18 Months; Test type: Superiority — Stratified Analysis; p = 0.0896, Cochran-Mantel-Haenszel; Difference in Proportion of Responders = 33.33, 95% CI 2-sided [-44.86 to 100.00]
Statistical Analysis 14: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Emotional Functioning, Post-Treatment Follow Up 24 Months; Test type: Superiority — Stratified Analysis; Difference in Proportion of Responders = 50.00, 95% CI 2-sided [-94.30 to 100.00]
Statistical Analysis 15: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Physical Functioning, Presurgical/Surgery; Test type: Superiority — Stratified Analysis; p = 0.7347, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.92, 95% CI 2-sided [0.56 to 1.50]
Statistical Analysis 16: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Physical Functioning, Cycle 4 Day 1; Test type: Superiority — Stratified Analysis; p = 0.0479, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.56, 95% CI 2-sided [0.32 to 1.00]
Statistical Analysis 17: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Physical Functioning, Cycle 6 Day 1; Test type: Superiority — Stratified Analysis; p = 0.0712, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.61, 95% CI 2-sided [0.36 to 1.05]
Statistical Analysis 18: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Physical Functioning, Cycle 8 Day 1; Test type: Superiority — Stratified Analysis; p = 0.8168, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.94, 95% CI 2-sided [0.56 to 1.58]
Statistical Analysis 19: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Physical Functioning, Cycle 12 Day 1; Test type: Superiority — Stratified Analysis; p = 0.6417, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.88, 95% CI 2-sided [0.50 to 1.52]
Statistical Analysis 20: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Physical Functioning, Cycle 16 Day 1; Test type: Superiority — Stratified Analysis; p = 0.8821, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.96, 95% CI 2-sided [0.53 to 1.72]
Statistical Analysis 21: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Physical Functioning, Cycle 20 Day 1; Test type: Superiority — Stratified Analysis; p = 0.2158, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.64, 95% CI 2-sided [0.32 to 1.30]
Statistical Analysis 22: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Physical Functioning, Completion of Treatment/Early Termination Visit; Test type: Superiority; p = 0.4762, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.84, 95% CI 2-sided [0.51 to 1.37]
Statistical Analysis 23: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Physical Functioning, Post-Treatment Follow Up 3 Months; Test type: Superiority — Stratified Analysis; p = 0.7585, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.10, 95% CI 2-sided [0.61 to 1.96]
Statistical Analysis 24: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Physical Functioning, Post-Treatment Follow Up 6 Months; Test type: Superiority — Stratified Analysis; p = 0.9985, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.00, 95% CI 2-sided [0.52 to 1.93]
Statistical Analysis 25: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Physical Functioning, Post-Treatment Follow Up 9 Months; Test type: Superiority — Stratified Analysis; p = 0.1067, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 2.07, 95% CI 2-sided [0.85 to 5.06]
Statistical Analysis 26: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Physical Functioning, Post-Treatment Follow Up 12 Months; Test type: Superiority — Stratified Analysis; p = 0.6171, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.42, 95% CI 2-sided [0.36 to 5.61]
Statistical Analysis 27: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Physical Functioning, Post-Treatment Follow Up 18 Months; Test type: Superiority — Stratified Analysis; p = 0.8084, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.41, 95% CI 2-sided [0.08 to 23.57]
Statistical Analysis 28: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Physical Functioning, Post-Treatment Follow Up 24 Months; Test type: Superiority — Stratified Analysis; p = 0.3173, Cochran-Mantel-Haenszel; Difference in Proportion of Responders = -50.00, 95% CI 2-sided [-100.00 to 94.30]
Statistical Analysis 29: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Global health status/QoL, Presurgical/Surgery; Test type: Superiority — Stratified Analysis; p = 0.6802, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.10, 95% CI 2-sided [0.69 to 1.77]
Statistical Analysis 30: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Global health status/QoL, Cycle 4 Day 1; Test type: Superiority — Stratified Analysis; p = 0.3470, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.79, 95% CI 2-sided [0.48 to 1.29]
Statistical Analysis 31: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Global health status/QoL, Cycle 6 Day 1; Test type: Superiority — Stratified Analysis; p = 0.5564, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.86, 95% CI 2-sided [0.53 to 1.41]
Statistical Analysis 32: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Global health status/QoL, Cycle 8 Day 1; Test type: Superiority — Stratified Analysis; p = 0.5000, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.19, 95% CI 2-sided [0.72 to 1.99]
Statistical Analysis 33: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Global health status/QoL, Cycle 12 Day 1; Test type: Superiority — Stratified Analysis; p = 0.9778, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.01, 95% CI 2-sided [0.57 to 1.78]
Statistical Analysis 34: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Global health status/QoL, Cycle 16 Day 1; Test type: Superiority — Stratified Analysis; p = 0.6005, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.17, 95% CI 2-sided [0.65 to 2.12]
Statistical Analysis 35: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Global health status/QoL, Cycle 20 Day 1; Test type: Superiority — Stratified Analysis; p = 0.9900, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.00, 95% CI 2-sided [0.50 to 2.00]
Statistical Analysis 36: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Global health status/QoL, Completion of Treatment/Early Termination Visit; Test type: Superiority — Stratified Analysis; p = 0.2634, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.32, 95% CI 2-sided [0.81 to 2.15]
Statistical Analysis 37: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Global health status/QoL, Post-Treatment Follow Up 3 Months; Test type: Superiority — Stratified Analysis; p = 0.9640, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.99, 95% CI 2-sided [0.56 to 1.74]
Statistical Analysis 38: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Global health status/QoL, Post-Treatment Follow Up 6 Months; Test type: Superiority — Stratified Analysis; p = 0.4117, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.76, 95% CI 2-sided [0.40 to 1.46]
Statistical Analysis 39: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Global health status/QoL, Post-Treatment Follow Up 9 Months; Test type: Superiority — Stratified Analysis; p = 0.3505, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.51, 95% CI 2-sided [0.63 to 3.62]
Statistical Analysis 40: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Global health status/QoL, Post-Treatment Follow Up 12 Months; Test type: Superiority — Stratified Analysis; p = 0.2439, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 2.28, 95% CI 2-sided [0.55 to 9.45]
Statistical Analysis 41: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Global health status/QoL, Post-Treatment Follow Up 18 Months; Test type: Superiority — Stratified Analysis; p = 0.1573, Cochran-Mantel-Haenszel; Difference in Proportion of Responders = 33.33, 95% CI 2-sided [-44.86 to 100.00]
Statistical Analysis 42: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Global health status/QoL, Post-Treatment Follow Up 24 Months; Test type: Superiority — Stratified Analysis; Difference in Proportion of Responders = 50.00, 95% CI 2-sided [-94.30 to 100.00]
Statistical Analysis 43: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Role Functioning, Presurgical/Surgery; Test type: Superiority — Stratified Analysis; p = 0.1820, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.72, 95% CI 2-sided [0.45 to 1.16]
Statistical Analysis 44: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Role functioning, Cycle 4 Day 1; Test type: Superiority — Stratified Analysis; p = 0.0046, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.47, 95% CI 2-sided [0.28 to 0.80]
Statistical Analysis 45: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Role functioning, Cycle 6 Day 1; Test type: Superiority — Stratified Analysis; p = 0.0361, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.59, 95% CI 2-sided [0.36 to 0.97]
Statistical Analysis 46: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Role functioning, Cycle 8 Day 1; Test type: Superiority — Stratified Analysis; p = 0.0848, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.64, 95% CI 2-sided [0.39 to 1.06]
Statistical Analysis 47: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Role functioning, Cycle 12 Day 1; Test type: Superiority — Stratified Analysis; p = 0.1224, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.64, 95% CI 2-sided [0.37 to 1.13]
Statistical Analysis 48: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Role functioning, Cycle 16 Day 1; Test type: Superiority — Stratified Analysis; p = 0.3127, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.74, 95% CI 2-sided [0.41 to 1.33]
Statistical Analysis 49: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Role functioning, Cycle 20 Day 1; Test type: Superiority — Stratified Analysis; p = 0.6065, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.84, 95% CI 2-sided [0.42 to 1.65]
Statistical Analysis 50: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Role functioning, Completion of Treatment/ Early Termination Visit; Test type: Superiority — Stratified Analysis; p = 0.2173, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.74, 95% CI 2-sided [0.45 to 1.20]
Statistical Analysis 51: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Role functioning, Post-Treatment Follow Up 3 Months; Test type: Superiority — Stratified Analysis; p = 0.1316, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.64, 95% CI 2-sided [0.35 to 1.15]
Statistical Analysis 52: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Role functioning, Post-Treatment Follow Up 6 Months; Test type: Superiority — Stratified Analysis; p = 0.7678, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.90, 95% CI 2-sided [0.46 to 1.76]
Statistical Analysis 53: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Role functioning, Post-Treatment Follow Up 9 Months; Test type: Superiority — Stratified Analysis; p = 0.7331, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.85, 95% CI 2-sided [0.34 to 2.14]
Statistical Analysis 54: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Role functioning, Post-Treatment Follow Up 12 Months; Test type: Superiority — Stratified Analysis; p = 0.1235, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 2.83, 95% CI 2-sided [0.73 to 10.92]
Statistical Analysis 55: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Role functioning, Post-Treatment Follow Up 18 Months; Test type: Superiority — Stratified Analysis; Difference in Proportion of Responders = 0.00, 95% CI 2-sided [-84.09 to 84.09]
Statistical Analysis 56: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Role functioning, Post-Treatment Follow Up 24 Months; Test type: Superiority — Stratified Analysis; Difference in Proportion of Responders = 50.00, 95% CI 2-sided [-94.30 to 100.00]
Statistical Analysis 57: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Social functioning, Presurgical/Surgery; Test type: Superiority — Stratified Analysis; p = 0.7869, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.07, 95% CI 2-sided [0.65 to 1.78]
Statistical Analysis 58: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Social functioning, Cycle 4 Day 1; Test type: Superiority — Stratified Analysis; p = 0.2502, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.73, 95% CI 2-sided [0.43 to 1.25]
Statistical Analysis 59: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Social functioning, Cycle 6 Day 1; Test type: Superiority — Stratified Analysis; p = 0.5066, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.84, 95% CI 2-sided [0.50 to 1.41]
Statistical Analysis 60: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Social functioning, Cycle 8 Day 1; Test type: Superiority — Stratified Analysis; p = 0.8124, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.94, 95% CI 2-sided [0.56 to 1.59]
Statistical Analysis 61: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Social functioning, Cycle 12 Day 1; Test type: Superiority — Stratified Analysis; p = 0.4656, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.23, 95% CI 2-sided [0.70 to 2.17]
Statistical Analysis 62: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Social functioning, Cycle 16 Day 1; Test type: Superiority — Stratified Analysis; p = 0.6725, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.14, 95% CI 2-sided [0.62 to 2.12]
Statistical Analysis 63: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Social functioning, Cycle 20 Day 1; Test type: Superiority — Stratified Analysis; p = 0.5780, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.82, 95% CI 2-sided [0.41 to 1.64]
Statistical Analysis 64: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Social functioning, Completion of Treatment/Early Termination Visit; Test type: Superiority — Stratified Analysis; p = 0.7611, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.08, 95% CI 2-sided [0.66 to 1.76]
Statistical Analysis 65: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Social functioning, Post-Treatment Follow Up 3 Months; Test type: Superiority — Stratified Analysis; p = 0.7588, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.09, 95% CI 2-sided [0.62 to 1.94]
Statistical Analysis 66: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Social functioning, Post-Treatment Follow Up 6 Months; Test type: Superiority — Stratified Analysis; p = 0.1428, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.60, 95% CI 2-sided [0.30 to 1.19]
Statistical Analysis 67: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Social functioning, Post-Treatment Follow Up 9 Months; Test type: Superiority — Stratified Analysis; p = 0.9802, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.99, 95% CI 2-sided [0.41 to 2.39]
Statistical Analysis 68: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Social functioning, Post-Treatment Follow Up 12 Months; Test type: Superiority — Stratified Analysis; p = 0.1967, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 2.34, 95% CI 2-sided [0.63 to 8.70]
Statistical Analysis 69: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Social functioning, Post-Treatment Follow Up 18 Months; Test type: Superiority — Stratified Analysis; p = 0.4795, Cochran-Mantel-Haenszel; Difference in Proportion of Respnders = 8.33, 95% CI 2-sided [-69.28 to 85.94]
Statistical Analysis 70: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Social functioning, Post-Treatment Follow Up 24 Months; Test type: Superiority — Stratified Analysis; Difference in Proportion of Responders = 50.00, 95% CI 2-sided [-94.30 to 100.00]

11. Secondary Outcome: Percentage of Participants Who Achieve a Clinically-Meaningful Improvement in Patient-Reported Function and HRQoL - Primary Tumor-Reductive Surgery Group
Description: Percentage of participants with clinical improvement, defined as >= 10-point increase from the baseline score on each of the functional (physical, role, emotional, and social) and GHS/QoL scales of the EORTC QLQ-C30.
Time Frame: as for outcome 9
Population: as for outcome 10
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo With Paclitaxel, Carboplatin and Bevacizumab | Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab
Number analyzed (Participants) | 473 | 473
Percentage of participants
  Physical Functioning, Cycle 3 Day 1: number analyzed (Participants) | 456 | 444
  Physical Functioning, Cycle 3 Day 1 | 22.6 | 19.8
  Physical Functioning, Cycle 5 Day 1: number analyzed (Participants) | 439 | 423
  Physical Functioning, Cycle 5 Day 1 | 23.7 | 21.3
  Physical Functioning, Cycle 8 Day 1: number analyzed (Participants) | 414 | 403
  Physical Functioning, Cycle 8 Day 1 | 28.7 | 27.0
  Physical Functioning, Cycle 12 Day 1: number analyzed (Participants) | 378 | 358
  Physical Functioning, Cycle 12 Day 1 | 35.4 | 32.4
  Physical Functioning, Cycle 16 Day 1: number analyzed (Participants) | 333 | 312
  Physical Functioning, Cycle 16 Day 1 | 32.1 | 34.3
  Physical Functioning, Cycle 20 Day 1: number analyzed (Participants) | 253 | 234
  Physical Functioning, Cycle 20 Day 1 | 34.8 | 32.5
  Physical Functioning, Completion of Treatment/Early Termination Visit: number analyzed (Participants) | 370 | 366
  Physical Functioning, Completion of Treatment/Early Termination Visit | 32.4 | 30.3
  Physical Functioning, Post-Treatment Follow Up 3 Months: number analyzed (Participants) | 235 | 236
  Physical Functioning, Post-Treatment Follow Up 3 Months | 35.7 | 28.4
  Physical Functioning, Post-Treatment Follow Up 6 Months: number analyzed (Participants) | 147 | 164
  Physical Functioning, Post-Treatment Follow Up 6 Months | 32.7 | 31.1
  Physical Functioning, Post-Treatment Follow Up 9 Months: number analyzed (Participants) | 84 | 98
  Physical Functioning, Post-Treatment Follow Up 9 Months | 34.5 | 27.6
  Physical Functioning, Post-Treatment Follow Up 12 Months: number analyzed (Participants) | 45 | 58
  Physical Functioning, Post-Treatment Follow Up 12 Months | 37.8 | 24.1
  Physical Functioning, Post-Treatment Follow Up 18 Months: number analyzed (Participants) | 14 | 16
  Physical Functioning, Post-Treatment Follow Up 18 Months | 42.9 | 18.8
  Physical Functioning, Post-Treatment Follow Up 24 Months: number analyzed (Participants) | 2 | 6
  Physical Functioning, Post-Treatment Follow Up 24 Months | 0 | 16.7
  Role Functioning, Cycle 3 Day 1: number analyzed (Participants) | 455 | 443
  Role Functioning, Cycle 3 Day 1 | 42.6 | 40.9
  Role Functioning, Cycle 5 Day 1: number analyzed (Participants) | 438 | 422
  Role Functioning, Cycle 5 Day 1 | 42.9 | 38.9
  Role Functioning, Cycle 8 Day 1: number analyzed (Participants) | 413 | 401
  Role Functioning, Cycle 8 Day 1 | 47.5 | 45.9
  Role Functioning, Cycle 12 Day 1: number analyzed (Participants) | 377 | 358
  Role Functioning, Cycle 12 Day 1 | 50.1 | 50.6
  Role Functioning, Cycle 16 Day 1: number analyzed (Participants) | 333 | 311
  Role Functioning, Cycle 16 Day 1 | 52.0 | 50.8
  Role Functioning, Cycle 20 Day 1: number analyzed (Participants) | 253 | 233
  Role Functioning, Cycle 20 Day 1 | 53.8 | 51.5
  Role Functioning, Completion of Treatment/ Early Termination Visit: number analyzed (Participants) | 370 | 367
  Role Functioning, Completion of Treatment/ Early Termination Visit | 48.4 | 46.6
  Role Functioning, Post-Treatment Follow Up 3 Months: number analyzed (Participants) | 235 | 236
  Role Functioning, Post-Treatment Follow Up 3 Months | 54.0 | 45.3
  Role Functioning, Post-Treatment Follow Up 6 Months: number analyzed (Participants) | 147 | 164
  Role Functioning, Post-Treatment Follow Up 6 Months | 55.1 | 43.9
  Role Functioning, Post-Treatment Follow Up 9 Months: number analyzed (Participants) | 84 | 98
  Role Functioning, Post-Treatment Follow Up 9 Months | 57.1 | 38.8
  Role Functioning, Post-Treatment Follow Up 12 Months: number analyzed (Participants) | 45 | 58
  Role Functioning, Post-Treatment Follow Up 12 Months | 60 | 27.6
  Role Functioning, Post-Treatment Follow Up 18 Months: number analyzed (Participants) | 14 | 16
  Role Functioning, Post-Treatment Follow Up 18 Months | 50 | 43.8
  Role Functioning, Post-Treatment Follow Up 24 Months: number analyzed (Participants) | 2 | 6
  Role Functioning, Post-Treatment Follow Up 24 Months | 50 | 16.7
  Social Functioning, Cycle 3 Day 1: number analyzed (Participants) | 455 | 442
  Social Functioning, Cycle 3 Day 1 | 30.1 | 31.4
  Social Functioning, Cycle 5 Day 1: number analyzed (Participants) | 439 | 422
  Social Functioning, Cycle 5 Day 1 | 32.6 | 32.0
  Social Functioning, Cycle 8 Day 1: number analyzed (Participants) | 413 | 403
  Social Functioning, Cycle 8 Day 1 | 37.8 | 38.7
  Social Functioning, Cycle 12 Day 1: number analyzed (Participants) | 376 | 357
  Social Functioning, Cycle 12 Day 1 | 42.6 | 41.2
  Social Functioning, Cycle 16 Day 1: number analyzed (Participants) | 333 | 312
  Social Functioning, Cycle 16 Day 1 | 43.5 | 48.7
  Social Functioning, Cycle 20 Day 1: number analyzed (Participants) | 252 | 234
  Social Functioning, Cycle 20 Day 1 | 45.6 | 50.0
  Social Functioning, Completion of Treatment/ Early Termination Visit: number analyzed (Participants) | 367 | 367
  Social Functioning, Completion of Treatment/ Early Termination Visit | 40.6 | 40.1
  Social Functioning, Post-Treatment Follow Up 3 Months: number analyzed (Participants) | 234 | 236
  Social Functioning, Post-Treatment Follow Up 3 Months | 42.7 | 41.1
  Social Functioning, Post-Treatment Follow Up 6 Months: number analyzed (Participants) | 148 | 164
  Social Functioning, Post-Treatment Follow Up 6 Months | 43.2 | 34.1
  Social Functioning, Post-Treatment Follow Up 9 Months: number analyzed (Participants) | 84 | 98
  Social Functioning, Post-Treatment Follow Up 9 Months | 50.0 | 36.7
  Social Functioning, Post-Treatment Follow Up 12 Months: number analyzed (Participants) | 45 | 58
  Social Functioning, Post-Treatment Follow Up 12 Months | 62.2 | 36.2
  Social Functioning, Post-Treatment Follow Up 18 Months: number analyzed (Participants) | 14 | 16
  Social Functioning, Post-Treatment Follow Up 18 Months | 57.1 | 43.8
  Social Functioning, Post-Treatment Follow Up 24 Months: number analyzed (Participants) | 2 | 6
  Social Functioning, Post-Treatment Follow Up 24 Months | 100 | 50.0
  Emotional Functioning, Cycle 3 Day 1: number analyzed (Participants) | 454 | 443
  Emotional Functioning, Cycle 3 Day 1 | 29.7 | 28.4
  Emotional Functioning, Cycle 5 Day 1: number analyzed (Participants) | 439 | 422
  Emotional Functioning, Cycle 5 Day 1 | 30.3 | 30.3
  Emotional Functioning, Cycle 8 Day 1: number analyzed (Participants) | 412 | 403
  Emotional Functioning, Cycle 8 Day 1 | 32.3 | 33.0
  Emotional Functioning, Cycle 12 Day 1: number analyzed (Participants) | 376 | 357
  Emotional Functioning, Cycle 12 Day 1 | 34.6 | 36.1
  Emotional Functioning, Cycle 16 Day 1: number analyzed (Participants) | 333 | 312
  Emotional Functioning, Cycle 16 Day 1 | 31.8 | 35.9
  Emotional Functioning, Cycle 20 Day 1: number analyzed (Participants) | 252 | 234
  Emotional Functioning, Cycle 20 Day 1 | 35.3 | 36.8
  Emotional Functioning, Completion of Treatment/ Early Termination Visit: number analyzed (Participants) | 368 | 367
  Emotional Functioning, Completion of Treatment/ Early Termination Visit | 27.7 | 28.6
  Emotional Functioning, Post-Treatment Follow Up 3 Months: number analyzed (Participants) | 234 | 236
  Emotional Functioning, Post-Treatment Follow Up 3 Months | 29.1 | 27.5
  Emotional Functioning, Post-Treatment Follow Up 6 Months: number analyzed (Participants) | 148 | 164
  Emotional Functioning, Post-Treatment Follow Up 6 Months | 30.4 | 37.8
  Emotional Functioning, Post-Treatment Follow Up 9 Months: number analyzed (Participants) | 84 | 98
  Emotional Functioning, Post-Treatment Follow Up 9 Months | 38.1 | 33.7
  Emotional Functioning, Post-Treatment Follow Up 12 Months: number analyzed (Participants) | 45 | 58
  Emotional Functioning, Post-Treatment Follow Up 12 Months | 44.4 | 34.5
  Emotional Functioning, Post-Treatment Follow Up 18 Months: number analyzed (Participants) | 14 | 16
  Emotional Functioning, Post-Treatment Follow Up 18 Months | 42.9 | 31.3
  Emotional Functioning, Post-Treatment Follow Up 24 Months: number analyzed (Participants) | 2 | 6
  Emotional Functioning, Post-Treatment Follow Up 24 Months | 50.0 | 16.7
  GHS/OoL, Cycle 3 Day 1: number analyzed (Participants) | 455 | 443
  GHS/OoL, Cycle 3 Day 1 | 32.3 | 34.5
  GHS/OoL, Cycle 5 Day 1: number analyzed (Participants) | 439 | 422
  GHS/OoL, Cycle 5 Day 1 | 33.0 | 31.0
  GHS/OoL, Cycle 8 Day 1: number analyzed (Participants) | 413 | 403
  GHS/OoL, Cycle 8 Day 1 | 39.5 | 38.7
  GHS/OoL, Cycle 12 Day 1: number analyzed (Participants) | 376 | 357
  GHS/OoL, Cycle 12 Day 1 | 41.5 | 43.4
  GHS/OoL, Cycle 16 Day 1: number analyzed (Participants) | 333 | 312
  GHS/OoL, Cycle 16 Day 1 | 42.9 | 42.9
  GHS/OoL, Cycle 20 Day 1: number analyzed (Participants) | 252 | 234
  GHS/OoL, Cycle 20 Day 1 | 42.5 | 46.2
  GHS/OoL, Completion of Treatment/ Early Termination Visit: number analyzed (Participants) | 368 | 367
  GHS/OoL, Completion of Treatment/ Early Termination Visit | 38.0 | 34.9
  GHS/OoL, Post-Treatment Follow Up 3 Months: number analyzed (Participants) | 234 | 236
  GHS/OoL, Post-Treatment Follow Up 3 Months | 40.6 | 38.6
  GHS/OoL, Post-Treatment Follow Up 6 Months: number analyzed (Participants) | 148 | 164
  GHS/OoL, Post-Treatment Follow Up 6 Months | 39.2 | 34.1
  GHS/OoL, Post-Treatment Follow Up 9 Months: number analyzed (Participants) | 84 | 98
  GHS/OoL, Post-Treatment Follow Up 9 Months | 39.3 | 35.7
  GHS/OoL, Post-Treatment Follow Up 12 Months: number analyzed (Participants) | 45 | 58
  GHS/OoL, Post-Treatment Follow Up 12 Months | 40.0 | 32.8
  GHS/OoL, Post-Treatment Follow Up 18 Months: number analyzed (Participants) | 14 | 16
  GHS/OoL, Post-Treatment Follow Up 18 Months | 42.9 | 18.8
  GHS/OoL, Post-Treatment Follow Up 24 Months: number analyzed (Participants) | 2 | 6
  GHS/OoL, Post-Treatment Follow Up 24 Months | 100 | 33.3
Statistical Analysis 1: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Emotional functioning, Cycle 3 Day 1; Test type: Superiority — Stratified Analysis; p = 0.6651, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.94, 95% CI 2-sided [0.70 to 1.25]
Statistical Analysis 2: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Emotional functioning, Cycle 5 Day 1; Test type: Superiority — Stratified Analysis; p = 0.9927, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.00, 95% CI 2-sided [0.75 to 1.34]
Statistical Analysis 3: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Emotional functioning, Cycle 8 Day 1; Test type: Superiority — Stratified Analysis; p = 0.8209, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.03, 95% CI 2-sided [0.77 to 1.39]
Statistical Analysis 4: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Emotional functioning, Cycle 12 Day 1; Test type: Superiority — Stratified Analysis; p = 0.6507, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.07, 95% CI 2-sided [0.79 to 1.45]
Statistical Analysis 5: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Emotional functioning, Cycle 16 Day 1; Test type: Superiority — Stratified Analysis; p = 0.2596, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.21, 95% CI 2-sided [0.87 to 1.67]
Statistical Analysis 6: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Emotional functioning, Cycle 20 Day 1; Test type: Superiority — Stratified Analysis; p = 0.6532, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.09, 95% CI 2-sided [0.75 to 1.58]
Statistical Analysis 7: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Emotional functioning, Completion Of Treatment/ Early Termination Visit; Test type: Superiority — Stratified Analysis; p = 0.7592, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.05, 95% CI 2-sided [0.76 to 1.45]
Statistical Analysis 8: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Emotional functioning, Post-Treatment Follow Up 3 Months; Test type: Superiority — Stratified Analysis; p = 0.7424, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.93, 95% CI 2-sided [0.62 to 1.40]
Statistical Analysis 9: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Emotional functioning, Post-Treatment Follow Up 6 Months; Test type: Superiority — Stratified Analysis; p = 0.1912, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.37, 95% CI 2-sided [0.85 to 2.19]
Statistical Analysis 10: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Emotional functioning, Post-Treatment Follow Up 9 Months; Test type: Superiority — Stratified Analysis; p = 0.5526, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.83, 95% CI 2-sided [0.45 to 1.53]
Statistical Analysis 11: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Emotional functioning, Post-Treatment Follow Up 12 Months; Test type: Superiority — Stratified Analysis; p = 0.3609, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.69, 95% CI 2-sided [0.32 to 1.52]
Statistical Analysis 12: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Emotional functioning, Post-Treatment Follow Up 18 Months; Test type: Superiority — Stratified Analysis; p = 0.7527, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.80, 95% CI 2-sided [0.20 to 3.23]
Statistical Analysis 13: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Emotional functioning, Post-Treatment Follow Up 24 Months; Test type: Superiority — Stratified Analysis; Difference in Proportion of Responders = -33.33, 95% CI 2-sided [-100.00 to 75.44]
Statistical Analysis 14: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Physical functioning, Cycle 3 Day 1; Test type: Superiority — Stratified Analysis; p = 0.3177, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.85, 95% CI 2-sided [0.62 to 1.17]
Statistical Analysis 15: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Physical functioning, Cycle 5 Day 1; Test type: Superiority — Stratified Analysis; p = 0.4184, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.88, 95% CI 2-sided [0.63 to 1.21]
Statistical Analysis 16: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Physical functioning, Cycle 8 Day 1; Test type: Superiority — Stratified Analysis; p = 0.5710, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.91, 95% CI 2-sided [0.67 to 1.24]
Statistical Analysis 17: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Physical functioning, Cycle 12 Day 1; Test type: Superiority — Stratified Analysis; p = 0.3973, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.88, 95% CI 2-sided [0.65 to 1.19]
Statistical Analysis 18: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Physical functioning, Cycle 16 Day 1; Test type: Superiority — Stratified Analysis; p = 0.5163, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.12, 95% CI 2-sided [0.80 to 1.55]
Statistical Analysis 19: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Physical functioning, Cycle 20 Day 1; Test type: Superiority — Stratified Analysis; p = 0.6897, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.93, 95% CI 2-sided [0.64 to 1.35]
Statistical Analysis 20: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Physical functioning, Completion Of Treatment/ Early Termination Visit; Test type: Superiority — Stratified Analysis; p = 0.5735, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.91, 95% CI 2-sided [0.67 to 1.25]
Statistical Analysis 21: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Physical functioning, Post-Treatment Follow Up 3 Months; Test type: Superiority — Stratified Analysis; p = 0.1414, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.75, 95% CI 2-sided [0.50 to 1.10]
Statistical Analysis 22: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Physical functioning, Post-Treatment Follow Up 6 Months; Test type: Superiority — Stratified Analysis; p = 0.8655, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.96, 95% CI 2-sided [0.59 to 1.55]
Statistical Analysis 23: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Physical functioning, Post-Treatment Follow Up 9 Months; Test type: Superiority — Stratified Analysis; p = 0.3017, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.72, 95% CI 2-sided [0.38 to 1.35]
Statistical Analysis 24: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Physical functioning, Post-Treatment Follow Up 12 Months; Test type: Superiority — Stratified Analysis; p = 0.2325, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.60, 95% CI 2-sided [0.26 to 1.39]
Statistical Analysis 25: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Physical functioning, Post-Treatment Follow Up 18 Months; Test type: Superiority — Stratified Analysis; p = 0.1717, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.33, 95% CI 2-sided [0.06 to 1.69]
Statistical Analysis 26: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Physical functioning, Post-Treatment Follow Up 24 Months; Test type: Superiority — Stratified Analsyis; Difference in Proportion of Responders = 16.67, 95% CI 2-sided [-46.49 to 79.82]
Statistical Analysis 27: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Global health status/QoL, Cycle 3 Day 1; Test type: Superiority — Stratified Analysis; p = 0.4745, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.11, 95% CI 2-sided [0.84 to 1.46]
Statistical Analysis 28: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Global health status/QoL, Cycle 5 Day 1; Test type: Superiority — Stratified Analysis; p = 0.5499, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.92, 95% CI 2-sided [0.69 to 1.22]
Statistical Analysis 29: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Global health status/QoL, Cycle 8 Day 1; Test type: Superiority — Stratified Analysis; p = 0.8436, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.97, 95% CI 2-sided [0.73 to 1.29]
Statistical Analysis 30: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Global health status/QoL, Cycle 12 Day 1; Test type: Superiority — Stratified Analysis; p = 0.5798, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.09, 95% CI 2-sided [0.81 to 1.46]
Statistical Analysis 31: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Global health status/QoL, Cycle 16 Day 1; Test type: Superiority — Stratified Analysis; p = 0.9094, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.02, 95% CI 2-sided [0.74 to 1.39]
Statistical Analysis 32: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Global health status/QoL, Cycle 20 Day 1; Test type: Superiority — Stratified Analysis; p = 0.4006, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.17, 95% CI 2-sided [0.81 to 1.67]
Statistical Analysis 33: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Global health status/QoL, Completion of Treatment/ Early Termination Visit; Test type: Superiority — Stratified Analysis; p = 0.4024, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.88, 95% CI 2-sided [0.65 to 1.19]
Statistical Analysis 34: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Global health status/QoL, Post-Treatment Follow Up 3 Months; Test type: Superiority — Stratified Analysis; p = 0.8796, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.97, 95% CI 2-sided [0.67 to 1.41]
Statistical Analysis 35: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Global health status/QoL, Post-Treatment Follow Up 6 Months; Test type: Superiority — Stratified Analysis; p = 0.4350, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.83, 95% CI 2-sided [0.53 to 1.32]
Statistical Analysis 36: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Global health status/QoL, Post-Treatment Follow Up 9 Months; Test type: Superiority — Stratified Analysis; p = 0.6225, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.86, 95% CI 2-sided [0.47 to 1.56]
Statistical Analysis 37: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Global health status/QoL, Post-Treatment Follow Up 12 Months; Test type: Superiority — Stratified Analysis; p = 0.5775, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.80, 95% CI 2-sided [0.36 to 1.77]
Statistical Analysis 38: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Global health status/QoL, Post-Treatment Follow Up 18 Months; Test type: Superiority — Stratified Analysis; p = 0.2343, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.37, 95% CI 2-sided [0.07 to 1.94]
Statistical Analysis 39: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Global health status/QoL, Post-Treatment Follow Up 24 Months; Test type: Superiority — Stratified Analysis; p = 0.0833, Cochran-Mantel-Haenszel; Difference in Proportion of Responders = -66.67, 95% CI 2-sided [-100.00 to 4.39]
Statistical Analysis 40: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Role functioning, Cycle 3 Day 1; Test type: Superiority — Superiority; p = 0.6012, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.93, 95% CI 2-sided [0.71 to 1.21]
Statistical Analysis 41: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Role functioning, Cycle 5 Day 1; Test type: Superiority — Stratified Analysis; p = 0.2291, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.85, 95% CI 2-sided [0.65 to 1.11]
Statistical Analysis 42: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Role functioning, Cycle 8 Day 1; Test type: Superiority — Stratified Analysis; p = 0.6574, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.94, 95% CI 2-sided [0.71 to 1.24]
Statistical Analysis 43: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Role functioning, Cycle 12 Day 1; Test type: Superiority — Stratified Analysis; p = 0.9217, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.01, 95% CI 2-sided [0.76 to 1.35]
Statistical Analysis 44: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Role functioning, Cycle 16 Day 1; Test type: Superiority — Stratified Analysis; p = 0.7693, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.95, 95% CI 2-sided [0.70 to 1.30]
Statistical Analysis 45: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Role functioning, Cycle 20 Day 1; Test type: Superiority — Stratified Analysis; p = 0.6470, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.92, 95% CI 2-sided [0.64 to 1.31]
Statistical Analysis 46: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Role functioning, Completion Of Treatment/ Early Termination Visit; Test type: Superiority — Stratified Analysis; p = 0.6391, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.93, 95% CI 2-sided [0.70 to 1.25]
Statistical Analysis 47: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Role functioning, Post-Treatment Follow Up 3 Months; Test type: Superiority — Stratified Analysis; p = 0.0892, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.73, 95% CI 2-sided [0.51 to 1.05]
Statistical Analysis 48: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Role functioning, Post-Treatment Follow Up 6 Months; Test type: Superiority — Stratified Analysis; p = 0.0550, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.65, 95% CI 2-sided [0.41 to 1.01]
Statistical Analysis 49: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Role functioning, Post-Treatment Follow Up 9 Months; Test type: Superiority — Stratified Analysis; p = 0.0168, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.49, 95% CI 2-sided [0.27 to 0.88]
Statistical Analysis 50: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Role functioning, Post-Treatment Follow Up 12 Months; Test type: Superiority — Stratified Analysis; p = 0.0021, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.29, 95% CI 2-sided [0.13 to 0.65]
Statistical Analysis 51: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Role functioning, Post-Treatment Follow Up 18 Months; Test type: Superiority — Stratified Analysis; p = 0.7817, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.80, 95% CI 2-sided [0.17 to 3.80]
Statistical Analysis 52: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Role functioning, Post-Treatment Follow Up 24 Months; Test type: Superiority — Stratified Analysis; Odds Ratio (OR) = -33.33, 95% CI 2-sided [-100.00 to 75.44]
Statistical Analysis 53: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Social functioning, Cycle 3 Day 1; Test type: Superiority — Stratified Analysis; p = 0.6646, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.06, 95% CI 2-sided [0.80 to 1.41]
Statistical Analysis 54: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Social functioning, Cycle 5 Day 1; Test type: Superiority — Stratified Analysis; p = 0.8677, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.98, 95% CI 2-sided [0.73 to 1.30]
Statistical Analysis 55: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Social functioning, Cycle 8 Day 1; Test type: Superiority — Stratified Analysis; p = 0.7670, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.04, 95% CI 2-sided [0.79 to 1.38]
Statistical Analysis 56: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Social functioning, Cycle 12 Day 1; Test type: Superiority; p = 0.7487, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.95, 95% CI 2-sided [0.71 to 1.28]
Statistical Analysis 57: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Social functioning, Cycle 16 Day 1; Test type: Superiority — Stratified Analysis; p = 0.1882, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.23, 95% CI 2-sided [0.90 to 1.68]
Statistical Analysis 58: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Social functioning, Cycle 20 Day 1; Test type: Superiority; p = 0.3015, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.21, 95% CI 2-sided [0.84 to 1.72]
Statistical Analysis 59: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Social functioning, Completion of Treatment/ Early Termination Visit; Test type: Superiority — Stratified Analysis; p = 0.9059, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.98, 95% CI 2-sided [0.73 to 1.32]
Statistical Analysis 60: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Social functioning, Post-Treatment Follow Up 3 Months; Test type: Superiority; p = 0.7125, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.93, 95% CI 2-sided [0.65 to 1.35]
Statistical Analysis 61: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Social functioning, Post-Treatment Follow Up 6 Months; Test type: Superiority — Stratified Analysis; p = 0.0947, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.68, 95% CI 2-sided [0.43 to 1.07]
Statistical Analysis 62: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Social functioning, Post-Treatment Follow Up 9 Months; Test type: Superiority — Stratified Analysis; p = 0.0686, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.58, 95% CI 2-sided [0.32 to 1.05]
Statistical Analysis 63: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Social functioning, Post-Treatment Follow Up 12 Months; Test type: Superiority — Stratified Analysis; p = 0.0175, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.39, 95% CI 2-sided [0.17 to 0.86]
Statistical Analysis 64: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Social functioning, Post-Treatment Follow Up 18 Months; Test type: Superiority — Stratified Analysis; p = 0.3376, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.46, 95% CI 2-sided [0.09 to 2.30]
Statistical Analysis 65: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Social functioning, Post-Treatment Follow Up 24 Months; Test type: Superiority; p = 0.5637, Cochran-Mantel-Haenszel; Difference in Proportion of Responders = -50.00, 95% CI 2-sided [-100.00 to 23.34]

12. Secondary Outcome: Percentage of Participants Who Remain Stable in Patient-Reported Function and HRQoL - Primary Tumor-Reductive Surgery Group
Description: Percentage of participants who remain stable defined as changes within 10 points from the baseline score on each of the functional (physical, role, emotional, and social) and GHS/QoL scales of the EORTC QLQ-C30.
Time Frame: as for outcome 9
Population: as for outcome 10
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo With Paclitaxel, Carboplatin and Bevacizumab | Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab
Number analyzed (Participants) | 473 | 473
Percentage of participants
  Physical Functioning, Cycle 3 Day 1: number analyzed (Participants) | 456 | 444
  Physical Functioning, Cycle 3 Day 1 | 53.1 | 56.1
  Physical Functioning, Cycle 5 Day 1: number analyzed (Participants) | 439 | 423
  Physical Functioning, Cycle 5 Day 1 | 49.0 | 50.1
  Physical Functioning, Cycle 8 Day 1: number analyzed (Participants) | 414 | 403
  Physical Functioning, Cycle 8 Day 1 | 47.8 | 49.4
  Physical Functioning, Cycle 12 Day 1: number analyzed (Participants) | 378 | 358
  Physical Functioning, Cycle 12 Day 1 | 47.1 | 51.1
  Physical Functioning, Cycle 16 Day 1: number analyzed (Participants) | 333 | 312
  Physical Functioning, Cycle 16 Day 1 | 50.5 | 48.7
  Physical Functioning, Cycle 20 Day 1: number analyzed (Participants) | 253 | 234
  Physical Functioning, Cycle 20 Day 1 | 46.6 | 50.9
  Physical Functioning, Completion of Treatment/ Early Termination Visit: number analyzed (Participants) | 370 | 366
  Physical Functioning, Completion of Treatment/ Early Termination Visit | 46.8 | 44.5
  Physical Functioning, Post-Treatment Follow Up 3 Months: number analyzed (Participants) | 235 | 236
  Physical Functioning, Post-Treatment Follow Up 3 Months | 41.3 | 47.9
  Physical Functioning, Post-Treatment Follow Up 6 Months: number analyzed (Participants) | 147 | 164
  Physical Functioning, Post-Treatment Follow Up 6 Months | 42.2 | 43.9
  Physical Functioning, Post-Treatment Follow Up 9 Months: number analyzed (Participants) | 84 | 98
  Physical Functioning, Post-Treatment Follow Up 9 Months | 46.4 | 46.9
  Physical Functioning, Post-Treatment Follow Up 12 Months: number analyzed (Participants) | 45 | 58
  Physical Functioning, Post-Treatment Follow Up 12 Months | 44.4 | 50.0
  Physical Functioning, Post-Treatment Follow Up 18 Months: number analyzed (Participants) | 14 | 16
  Physical Functioning, Post-Treatment Follow Up 18 Months | 35.7 | 56.3
  Physical Functioning, Post-Treatment Follow Up 24 Months: number analyzed (Participants) | 2 | 6
  Physical Functioning, Post-Treatment Follow Up 24 Months | 100 | 33.3
  Role Functioning, Cycle 3 Day 1: number analyzed (Participants) | 455 | 443
  Role Functioning, Cycle 3 Day 1 | 35.8 | 30.9
  Role Functioning, Cycle 5 Day 1: number analyzed (Participants) | 438 | 422
  Role Functioning, Cycle 5 Day 1 | 30.1 | 33.6
  Role Functioning, Cycle 8 Day 1: number analyzed (Participants) | 413 | 401
  Role Functioning, Cycle 8 Day 1 | 31.2 | 30.9
  Role Functioning, Cycle 12 Day 1: number analyzed (Participants) | 377 | 358
  Role Functioning, Cycle 12 Day 1 | 32.9 | 32.1
  Role Functioning, Cycle 16 Day 1: number analyzed (Participants) | 333 | 311
  Role Functioning, Cycle 16 Day 1 | 27.6 | 33.4
  Role Functioning, Cycle 20 Day 1: number analyzed (Participants) | 253 | 233
  Role Functioning, Cycle 20 Day 1 | 27.3 | 34.8
  Role Functioning, Completion of Treatment/ Early Termination Visit: number analyzed (Participants) | 370 | 367
  Role Functioning, Completion of Treatment/ Early Termination Visit | 28.6 | 28.6
  Role Functioning, Post-Treatment Follow Up 3 Months: number analyzed (Participants) | 235 | 236
  Role Functioning, Post-Treatment Follow Up 3 Months | 25.1 | 27.1
  Role Functioning, Post-Treatment Follow Up 6 Months: number analyzed (Participants) | 147 | 164
  Role Functioning, Post-Treatment Follow Up 6 Months | 24.5 | 29.9
  Role Functioning, Post-Treatment Follow Up 9 Months: number analyzed (Participants) | 84 | 98
  Role Functioning, Post-Treatment Follow Up 9 Months | 23.8 | 34.7
  Role Functioning, Post-Treatment Follow Up 12 Months: number analyzed (Participants) | 45 | 58
  Role Functioning, Post-Treatment Follow Up 12 Months | 33.3 | 34.5
  Role Functioning, Post-Treatment Follow Up 18 Months: number analyzed (Participants) | 14 | 16
  Role Functioning, Post-Treatment Follow Up 18 Months | 42.9 | 25.0
  Role Functioning, Post-Treatment Follow Up 24 Months: number analyzed (Participants) | 2 | 6
  Role Functioning, Post-Treatment Follow Up 24 Months | 50 | 66.7
  Social Functioning, Cycle 3 Day 1: number analyzed (Participants) | 455 | 442
  Social Functioning, Cycle 3 Day 1 | 40.7 | 36.7
  Social Functioning, Cycle 5 Day 1: number analyzed (Participants) | 439 | 422
  Social Functioning, Cycle 5 Day 1 | 37.6 | 36.7
  Social Functioning, Cycle 8 Day 1: number analyzed (Participants) | 413 | 403
  Social Functioning, Cycle 8 Day 1 | 40.2 | 35.2
  Social Functioning, Cycle 12 Day 1: number analyzed (Participants) | 376 | 357
  Social Functioning, Cycle 12 Day 1 | 38.3 | 39.2
  Social Functioning, Cycle 16 Day 1: number analyzed (Participants) | 333 | 312
  Social Functioning, Cycle 16 Day 1 | 36.6 | 33.3
  Social Functioning, Cycle 20 Day 1: number analyzed (Participants) | 252 | 234
  Social Functioning, Cycle 20 Day 1 | 34.1 | 33.8
  Social Functioning, Completion of Treatment/ Early Termination Visit: number analyzed (Participants) | 367 | 367
  Social Functioning, Completion of Treatment/ Early Termination Visit | 31.9 | 31.1
  Social Functioning, Post-Treatment Follow Up 3 Months: number analyzed (Participants) | 234 | 236
  Social Functioning, Post-Treatment Follow Up 3 Months | 30.3 | 32.6
  Social Functioning, Post-Treatment Follow Up 6 Months: number analyzed (Participants) | 148 | 164
  Social Functioning, Post-Treatment Follow Up 6 Months | 33.8 | 34.8
  Social Functioning, Post-Treatment Follow Up 9 Months: number analyzed (Participants) | 84 | 98
  Social Functioning, Post-Treatment Follow Up 9 Months | 27.4 | 30.6
  Social Functioning, Post-Treatment Follow Up 12 Months: number analyzed (Participants) | 45 | 58
  Social Functioning, Post-Treatment Follow Up 12 Months | 28.9 | 25.9
  Social Functioning, Post-Treatment Follow Up 18 Months: number analyzed (Participants) | 14 | 16
  Social Functioning, Post-Treatment Follow Up 18 Months | 28.6 | 18.8
  Social Functioning, Post-Treatment Follow Up 24 Months: number analyzed (Participants) | 2 | 6
  Social Functioning, Post-Treatment Follow Up 24 Months | 0 | 16.7
  Emotional Functioning, Cycle 3 Day 1: number analyzed (Participants) | 454 | 443
  Emotional Functioning, Cycle 3 Day 1 | 57.5 | 57.3
  Emotional Functioning, Cycle 5 Day 1: number analyzed (Participants) | 439 | 422
  Emotional Functioning, Cycle 5 Day 1 | 52.4 | 53.6
  Emotional Functioning, Cycle 8 Day 1: number analyzed (Participants) | 412 | 403
  Emotional Functioning, Cycle 8 Day 1 | 53.2 | 54.6
  Emotional Functioning, Cycle 12 Day 1: number analyzed (Participants) | 376 | 357
  Emotional Functioning, Cycle 12 Day 1 | 53.2 | 50.1
  Emotional Functioning, Cycle 16 Day 1: number analyzed (Participants) | 333 | 312
  Emotional Functioning, Cycle 16 Day 1 | 55.0 | 51.3
  Emotional Functioning, Cycle 20 Day 1: number analyzed (Participants) | 252 | 234
  Emotional Functioning, Cycle 20 Day 1 | 49.2 | 52.1
  Emotional Functioning, Completion of Treatment/ Early Termination Visit: number analyzed (Participants) | 368 | 367
  Emotional Functioning, Completion of Treatment/ Early Termination Visit | 53.0 | 51.8
  Emotional Functioning, Post-Treatment Follow Up 3 Months: number analyzed (Participants) | 234 | 236
  Emotional Functioning, Post-Treatment Follow Up 3 Months | 51.3 | 55.5
  Emotional Functioning, Post-Treatment Follow Up 6 Months: number analyzed (Participants) | 148 | 164
  Emotional Functioning, Post-Treatment Follow Up 6 Months | 48.6 | 47.6
  Emotional Functioning, Post-Treatment Follow Up 9 Months: number analyzed (Participants) | 84 | 98
  Emotional Functioning, Post-Treatment Follow Up 9 Months | 53.6 | 48.0
  Emotional Functioning, Post-Treatment Follow Up 12 Months: number analyzed (Participants) | 45 | 58
  Emotional Functioning, Post-Treatment Follow Up 12 Months | 46.7 | 43.1
  Emotional Functioning, Post-Treatment Follow Up 18 Months: number analyzed (Participants) | 14 | 16
  Emotional Functioning, Post-Treatment Follow Up 18 Months | 50.0 | 37.5
  Emotional Functioning, Post-Treatment Follow Up 24 Months: number analyzed (Participants) | 2 | 6
  Emotional Functioning, Post-Treatment Follow Up 24 Months | 50.0 | 16.7
  GHS/OoL, Cycle 3 Day 1: number analyzed (Participants) | 455 | 443
  GHS/OoL, Cycle 3 Day 1 | 43.3 | 42.2
  GHS/OoL, Cycle 5 Day 1: number analyzed (Participants) | 439 | 422
  GHS/OoL, Cycle 5 Day 1 | 42.6 | 44.8
  GHS/OoL, Cycle 8 Day 1: number analyzed (Participants) | 413 | 403
  GHS/OoL, Cycle 8 Day 1 | 39.0 | 42.9
  GHS/OoL, Cycle 12 Day 1: number analyzed (Participants) | 376 | 357
  GHS/OoL, Cycle 12 Day 1 | 40.7 | 42.9
  GHS/OoL, Cycle 16 Day 1: number analyzed (Participants) | 333 | 312
  GHS/OoL, Cycle 16 Day 1 | 38.4 | 43.3
  GHS/OoL, Cycle 20 Day 1: number analyzed (Participants) | 252 | 234
  GHS/OoL, Cycle 20 Day 1 | 36.9 | 42.3
  GHS/OoL, Completion of Treatment/ Early Termination Visit: number analyzed (Participants) | 368 | 367
  GHS/OoL, Completion of Treatment/ Early Termination Visit | 37.2 | 40.3
  GHS/OoL, Post-Treatment Follow Up 3 Months: number analyzed (Participants) | 234 | 236
  GHS/OoL, Post-Treatment Follow Up 3 Months | 38.9 | 38.6
  GHS/OoL, Post-Treatment Follow Up 6 Months: number analyzed (Participants) | 148 | 164
  GHS/OoL, Post-Treatment Follow Up 6 Months | 39.9 | 42.1
  GHS/OoL, Post-Treatment Follow Up 9 Months: number analyzed (Participants) | 84 | 98
  GHS/OoL, Post-Treatment Follow Up 9 Months | 39.3 | 38.8
  GHS/OoL, Post-Treatment Follow Up 12 Months: number analyzed (Participants) | 45 | 58
  GHS/OoL, Post-Treatment Follow Up 12 Months | 42.2 | 32.8
  GHS/OoL, Post-Treatment Follow Up 18 Months: number analyzed (Participants) | 14 | 16
  GHS/OoL, Post-Treatment Follow Up 18 Months | 35.7 | 37.5
  GHS/OoL, Post-Treatment Follow Up 24 Months: number analyzed (Participants) | 2 | 6
  GHS/OoL, Post-Treatment Follow Up 24 Months | 0 | 16.7
Statistical Analysis 1: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Emotional Functioning, Cycle 3 Day 1; Test type: Superiority — Stratified Analysis; p = 0.9770, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.00, 95% CI 2-sided [0.76 to 1.30]
Statistical Analysis 2: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Emotional Functioning, Cycle 5 Day 1; Test type: Superiority — Stratified Analysis; p = 0.7317, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.05, 95% CI 2-sided [0.80 to 1.37]
Statistical Analysis 3: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Emotional Functioning, Cycle 8 Day 1; Test type: Superiority; p = 0.6937, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.06, 95% CI 2-sided [0.80 to 1.39]
Statistical Analysis 4: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Emotional Functioning, Cycle 12 Day 1; Test type: Superiority — Stratified Analysis; p = 0.3916, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.88, 95% CI 2-sided [0.66 to 1.18]
Statistical Analysis 5: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Emotional Functioning, Cycle 16 Day 1; Test type: Superiority — Stratified Analysis; p = 0.3363, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.86, 95% CI 2-sided [0.63 to 1.17]
Statistical Analysis 6: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Emotional Functioning, Cycle 20 Day 1; Test type: Superiority; p = 0.6761, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.08, 95% CI 2-sided [0.75 to 1.55]
Statistical Analysis 7: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Emotional Functioning, Completion of Treatment/ Early Termination Visit; Test type: Superiority — Stratified Analysis; p = 0.6997, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.94, 95% CI 2-sided [0.71 to 1.26]
Statistical Analysis 8: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Emotional Functioning, Post-Treatment Follow Up 3 Months; Test type: Superiority — Stratified Analysis; p = 0.3592, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.19, 95% CI 2-sided [0.82 to 1.72]
Statistical Analysis 9: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Emotional Functioning, Post-Treatment Follow Up 6 Months; Test type: Superiority — Stratified Analysis; p = 0.8798, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.97, 95% CI 2-sided [0.62 to 1.51]
Statistical Analysis 10: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Emotional Functioning, Post-Treatment Follow Up 9 Months; Test type: Superiority — Stratified Analysis; p = 0.3857, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.77, 95% CI 2-sided [0.43 to 1.39]
Statistical Analysis 11: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Emotional Functioning, Post-Treatment Follow Up 12 Months; Test type: Superiority — Stratified Analysis; p = 0.6854, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.85, 95% CI 2-sided [0.39 to 1.85]
Statistical Analysis 12: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Emotional Functioning, Post-Treatment Follow Up 18 Months; Test type: Superiority — Stratified Analysis; p = 0.4533, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.54, 95% CI 2-sided [0.11 to 2.70]
Statistical Analysis 13: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Emotional Functioning, Post-Treatment Follow Up 24 Months; Test type: Superiority — Stratified Analysis; p = 0.3173, Cochran-Mantel-Haenszel; Difference in Proportion of Responders = -33.33, 95% CI 2-sided [-100.00 to 75.44]
Statistical Analysis 14: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Physical functioning, Cycle 3 Day 1; Test type: Superiority — Stratified Analysis; p = 0.3658, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.13, 95% CI 2-sided [0.87 to 1.47]
Statistical Analysis 15: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Physical functioning, Cycle 5 Day 1; Test type: Superiority — Stratified Analysis; p = 0.7619, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.04, 95% CI 2-sided [0.80 to 1.36]
Statistical Analysis 16: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Physical functioning, Cycle 8 Day 1; Test type: Superiority — Stratified Analysis; p = 0.6580, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.06, 95% CI 2-sided [0.81 to 1.40]
Statistical Analysis 17: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Physical functioning, Cycle 12 Day 1; Test type: Superiority — Stratified Analysis; p = 0.2726, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.18, 95% CI 2-sided [0.88 to 1.57]
Statistical Analysis 18: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Physical functioning, Cycle 16 Day 1; Test type: Superiority — Stratified Analysis; p = 0.6973, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.94, 95% CI 2-sided [0.69 to 1.29]
Statistical Analysis 19: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Physical functioning, Cycle 20 Day 1; Test type: Superiority — Stratified Analysis; p = 0.4470, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.15, 95% CI 2-sided [0.80 to 1.64]
Statistical Analysis 20: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Physical functioning, Completion of Treatment/ Early Termination Visit; Test type: Superiority — Stratified Analysis; p = 0.5150, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.91, 95% CI 2-sided [0.68 to 1.21]
Statistical Analysis 21: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Physical functioning, Post-Treatment Follow Up 3 Months; Test type: Superiority — Stratified Analysis; p = 0.2103, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.26, 95% CI 2-sided [0.88 to 1.82]
Statistical Analysis 22: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Physical functioning, Post-Treatment Follow Up 6 Months; Test type: Superiority — Stratified Analysis; p = 0.7969, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.06, 95% CI 2-sided [0.68 to 1.66]
Statistical Analysis 23: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Physical functioning, Post-Treatment Follow Up 9 Months; Test type: Superiority — Stratified Analysis; p = 0.8300, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.07, 95% CI 2-sided [0.60 to 1.91]
Statistical Analysis 24: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Physical functioning, Post-Treatment Follow Up 12 Months; Test type: Superiority — Stratified Analysis; p = 0.6987, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.17, 95% CI 2-sided [0.53 to 2.55]
Statistical Analysis 25: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Physical functioning, Post-Treatment Follow Up 18 Months; Test type: Superiority — Stratified Analysis; p = 0.1441, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 3.32, 95% CI 2-sided [0.62 to 17.77]
Statistical Analysis 26: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Physical functioning, Post-Treatment Follow Up 24 Months; Test type: Superiority — Stratified Analysis; p = 0.3173, Cochran-Mantel-Haenszel; Difference in proportion of Responders = -66.67, 95% CI 2-sided [-100.00 to 4.39]
Statistical Analysis 27: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Global health status/ QoL, Cycle 3 Day 1; Test type: Superiority — Stratified Analysis; p = 0.7591, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.96, 95% CI 2-sided [0.74 to 1.25]
Statistical Analysis 28: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Global health status/ QoL, Cycle 5 Day 1; Test type: Superiority — Stratified Analysis; p = 0.5403, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.09, 95% CI 2-sided [0.83 to 1.42]
Statistical Analysis 29: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Global health status/ QoL, Cycle 8 Day 1; Test type: Superiority — Stratified Analysis; p = 0.2654, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.17, 95% CI 2-sided [0.89 to 1.55]
Statistical Analysis 30: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Global health status/ QoL, Cycle 12 Day 1; Test type: Superiority; p = 0.5138, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.10, 95% CI 2-sided [0.82 to 1.48]
Statistical Analysis 31: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Global health status/ QoL, Cycle 16 Day 1; Test type: Superiority — Stratified Analysis; p = 0.2138, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.22, 95% CI 2-sided [0.89 to 1.67]
Statistical Analysis 32: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Global health status/ QoL, Cycle 20 Day 1; Test type: Superiority — Stratified Analysis; p = 0.2114, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.26, 95% CI 2-sided [0.88 to 1.82]
Statistical Analysis 33: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Global health status/ QoL, Completion of Treatment/ Early Termination Visit; Test type: Superiority — Stratified Analysis; p = 0.3938, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.14, 95% CI 2-sided [0.85 to 1.53]
Statistical Analysis 34: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Global health status/ QoL, Post-Treatment Follow Up 3 Months; Test type: Superiority — Stratified Analysis; p = 0.7793, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.95, 95% CI 2-sided [0.65 to 1.38]
Statistical Analysis 35: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Global health status/ QoL, Post-Treatment Follow Up 6 Months; Test type: Superiority — Stratified Analysis; p = 0.7370, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.08, 95% CI 2-sided [0.69 to 1.39]
Statistical Analysis 36: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Global health status/ QoL, Post-Treatment Follow Up 9 Months; Test type: Superiority — Stratified Analysis; p = 0.9658, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.99, 95% CI 2-sided [0.55 to 1.79]
Statistical Analysis 37: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Global health status/ QoL, Post-Treatment Follow Up 12 Months; Test type: Superiority — Stratified Analysis; p = 0.3015, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.66, 95% CI 2-sided [0.29 to 1.46]
Statistical Analysis 38: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Global health status/ QoL, Post-Treatment Follow Up 18 Months; Test type: Superiority — Stratified Analysis; p = 0.7534, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.77, 95% CI 2-sided [0.15 to 3.94]
Statistical Analysis 39: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Global health status/ QoL, Post-Treatment Follow Up 24 Months; Test type: Superiority — Stratified Analysis; p = 0.5637, Cochran-Mantel-Haenszel; Difference in Proportion of Responders = 16.67, 95% CI 2-sided [-46.49 to 79.82]
Statistical Analysis 40: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Role functioning, Cycle 3 Day 1; Test type: Superiority — Stratified Analysis; p = 0.1177, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.80, 95% CI 2-sided [0.61 to 1.06]
Statistical Analysis 41: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Role functioning, Cycle 5 Day 1; Test type: Superiority — Stratified Analysis; p = 0.2730, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.17, 95% CI 2-sided [0.88 to 1.56]
Statistical Analysis 42: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Role functioning, Cycle 8 Day 1; Test type: Superiority — Stratified Analysis; p = 0.9306, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.99, 95% CI 2-sided [0.73 to 1.33]
Statistical Analysis 43: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Role functioning, Cycle 12 Day 1; Test type: Superiority — Stratified Analysis; p = 0.8631, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.97, 95% CI 2-sided [0.72 to 1.32]
Statistical Analysis 44: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Role functioning, Cycle 16 Day 1; Test type: Superiority — Stratified Analysis; p = 0.0977, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.33, 95% CI 2-sided [0.95 to 1.86]
Statistical Analysis 45: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Role functioning, Cycle 20 Day 1; Test type: Superiority — Stratified Analysis; p = 0.0726, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.43, 95% CI 2-sided [0.97 to 2.10]
Statistical Analysis 46: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Role functioning, Completion of Treatment/ Early Termination Visit; Test type: Superiority — Stratified Analysis; p = 0.9974, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.00, 95% CI 2-sided [0.73 to 1.38]
Statistical Analysis 47: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Role functioning, Post-Treatment Follow Up 3 Months; Test type: Superiority — Stratified Analysis; p = 0.7069, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.08, 95% CI 2-sided [0.72 to 1.63]
Statistical Analysis 48: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Role functioning, Post-Treatment Follow Up 6 Months; Test type: Superiority — Stratified Analysis; p = 0.3068, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.30, 95% CI 2-sided [0.78 to 2.16]
Statistical Analysis 49: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Role functioning, Post-Treatment Follow Up 9 Months; Test type: Superiority — Stratified Analysis; p = 0.1375, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.64, 95% CI 2-sided [0.85 to 3.16]
Statistical Analysis 50: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Role functioning, Post-Treatment Follow Up 12 Months; Test type: Superiority — Stratified Analysis; p = 0.9540, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.02, 95% CI 2-sided [0.46 to 2.29]
Statistical Analysis 51: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Role functioning, Post-Treatment Follow Up 18 Months; Test type: Superiority — Stratified Analysis; p = 0.4283, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.53, 95% CI 2-sided [0.10 to 2.64]
Statistical Analysis 52: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Role functioning, Post-Treatment Follow Up 24 Months; Test type: Superiority — Stratified Analysis; Difference in Proportion of Responders = 16.67, 95% CI 2-sided [-95.56 to 100.00]
Statistical Analysis 53: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Social Functioning, Cycle 3 Day 1; Test type: Superiority — Stratified Analysis; p = 0.2153, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.84, 95% CI 2-sided [0.64 to 1.10]
Statistical Analysis 54: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Social Functioning, Cycle 5 Day 1; Test type: Superiority — Stratified Analysis; p = 0.7878, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.96, 95% CI 2-sided [0.73 to 1.27]
Statistical Analysis 55: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Social Functioning, Cycle 8 Day 1; Test type: Superiority — Stratified Analysis; p = 0.1544, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.81, 95% CI 2-sided [0.61 to 1.08]
Statistical Analysis 56: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Social Functioning, Cycle 12 Day 1; Test type: Superiority — Stratified Analysis; p = 0.8017, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.04, 95% CI 2-sided [0.77 to 1.40]
Statistical Analysis 57: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Social Functioning, Cycle 16 Day 1; Test type: Superiority — Stratified Analysis; p = 0.4295, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.88, 95% CI 2-sided [0.63 to 1.21]
Statistical Analysis 58: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Social Functioning, Cycle 20 Day 1; Test type: Superiority — Stratified Analysis; p = 0.9540, Cochran-Mantel-Haenszel; Odds Ratio, log = 0.99, 95% CI 2-sided [0.68 to 1.44]
Statistical Analysis 59: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Social Functioning, Completion of Treatment/ Early Termination Visit; Test type: Superiority — Stratified Analysis; p = 0.7494, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.95, 95% CI 2-sided [0.69 to 1.30]
Statistical Analysis 60: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Social Functioning, Post-Treatment Follow Up 3 Months; Test type: Superiority — Stratified Analysis; p = 0.6412, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.10, 95% CI 2-sided [0.74 to 1.62]
Statistical Analysis 61: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Social Functioning, Post-Treatment Follow Up 6 Months; Test type: Superiority — Stratified Analysis; p = 0.8652, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.04, 95% CI 2-sided [0.65 to 1.67]
Statistical Analysis 62: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Social Functioning, Post-Treatment Follow Up 9 Months; Test type: Superiority — Stratified Analysis; p = 0.6912, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.14, 95% CI 2-sided [0.60 to 2.18]
Statistical Analysis 63: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Social Functioning, Post-Treatment Follow Up 12 Months; Test type: Superiority — Stratified Analysis; p = 0.5834, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.79, 95% CI 2-sided [0.33 to 1.86]
Statistical Analysis 64: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Social Functioning, Post-Treatment Follow Up 18 Months; Test type: Superiority — Stratified Analysis; p = 0.9578, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.93, 95% CI 2-sided [0.05 to 16.05]
Statistical Analysis 65: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Social Functioning, Post-Treatment Follow Up 24 Months; Test type: Superiority — Stratified Analysis; p = 0.5637, Cochran-Mantel-Haenszel; Difference in Proportion of Responders = 16.67, 95% CI 2-sided [-46.49 to 79.82]

13. Secondary Outcome: Percentage of Participants With Deterioration in Patient-Reported Function and HRQoL - Primary Tumor-Reductive Surgery Group
Description: Percentage of participants with deterioration in patient-reported function and HRQoL, defined as >= 10 points decrease from the baseline score on each of the functional (physical, role, emotional, and social) and GHS/QoL scales of the EORTC QLQ-C30.
Time Frame: From randomization to the end of treatment/discontinuation (up to approximately 66 weeks), and during follow-up period (up to approximately 60 months). Cycle length=21 days.
Population: as for outcome 10
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo With Paclitaxel, Carboplatin and Bevacizumab | Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab
Number analyzed (Participants) | 473 | 473
Percentage of participants
  Physical Functioning, Cycle 3 Day 1: number analyzed (Participants) | 456 | 444
  Physical Functioning, Cycle 3 Day 1 | 24.1 | 24.1
  Physical Functioning, Cycle 5 Day 1: number analyzed (Participants) | 439 | 423
  Physical Functioning, Cycle 5 Day 1 | 27.1 | 28.6
  Physical Functioning, Cycle 8 Day 1: number analyzed (Participants) | 414 | 403
  Physical Functioning, Cycle 8 Day 1 | 23.4 | 23.6
  Physical Functioning, Cycle 12 Day 1: number analyzed (Participants) | 378 | 358
  Physical Functioning, Cycle 12 Day 1 | 17.2 | 16.5
  Physical Functioning, Cycle 16 Day 1: number analyzed (Participants) | 333 | 312
  Physical Functioning, Cycle 16 Day 1 | 17.1 | 17.0
  Physical Functioning, Cycle 20 Day 1: number analyzed (Participants) | 253 | 234
  Physical Functioning, Cycle 20 Day 1 | 18.2 | 16.7
  Physical Functioning, Completion of Treatment/ Early Termination Visit: number analyzed (Participants) | 370 | 366
  Physical Functioning, Completion of Treatment/ Early Termination Visit | 20.5 | 25.1
  Physical Functioning, Post-Treatment Follow Up 3 Months: number analyzed (Participants) | 235 | 236
  Physical Functioning, Post-Treatment Follow Up 3 Months | 22.6 | 23.7
  Physical Functioning, Post-Treatment Follow Up 6 Months: number analyzed (Participants) | 147 | 164
  Physical Functioning, Post-Treatment Follow Up 6 Months | 24.5 | 25.0
  Physical Functioning, Post-Treatment Follow Up 9 Months: number analyzed (Participants) | 84 | 98
  Physical Functioning, Post-Treatment Follow Up 9 Months | 19.0 | 25.5
  Physical Functioning, Post-Treatment Follow Up 12 Months: number analyzed (Participants) | 45 | 58
  Physical Functioning, Post-Treatment Follow Up 12 Months | 17.8 | 25.9
  Physical Functioning, Post-Treatment Follow Up 18 Months: number analyzed (Participants) | 14 | 16
  Physical Functioning, Post-Treatment Follow Up 18 Months | 21.4 | 25.0
  Physical Functioning, Post-Treatment Follow Up 24 Months: number analyzed (Participants) | 2 | 6
  Physical Functioning, Post-Treatment Follow Up 24 Months | 0 | 50
  Role Functioning, Cycle 3 Day 1: number analyzed (Participants) | 455 | 443
  Role Functioning, Cycle 3 Day 1 | 21.3 | 27.8
  Role Functioning, Cycle 5 Day 1: number analyzed (Participants) | 438 | 422
  Role Functioning, Cycle 5 Day 1 | 26.7 | 27.0
  Role Functioning, Cycle 8 Day 1: number analyzed (Participants) | 413 | 401
  Role Functioning, Cycle 8 Day 1 | 21.1 | 22.7
  Role Functioning, Cycle 12 Day 1: number analyzed (Participants) | 377 | 358
  Role Functioning, Cycle 12 Day 1 | 16.7 | 16.8
  Role Functioning, Cycle 16 Day 1: number analyzed (Participants) | 333 | 311
  Role Functioning, Cycle 16 Day 1 | 20.1 | 15.8
  Role Functioning, Cycle 20 Day 1: number analyzed (Participants) | 253 | 233
  Role Functioning, Cycle 20 Day 1 | 18.6 | 13.3
  Role Functioning, Completion of Treatment/ Early Termination Visit: number analyzed (Participants) | 370 | 367
  Role Functioning, Completion of Treatment/ Early Termination Visit | 23.0 | 24.3
  Role Functioning, Post-Treatment Follow Up 3 Months: number analyzed (Participants) | 235 | 236
  Role Functioning, Post-Treatment Follow Up 3 Months | 20.9 | 27.1
  Role Functioning, Post-Treatment Follow Up 6 Months: number analyzed (Participants) | 147 | 164
  Role Functioning, Post-Treatment Follow Up 6 Months | 20.4 | 25.6
  Role Functioning, Post-Treatment Follow Up 9 Months: number analyzed (Participants) | 84 | 98
  Role Functioning, Post-Treatment Follow Up 9 Months | 19.0 | 26.5
  Role Functioning, Post-Treatment Follow Up 12 Months: number analyzed (Participants) | 45 | 58
  Role Functioning, Post-Treatment Follow Up 12 Months | 6.7 | 37.9
  Role Functioning, Post-Treatment Follow Up 18 Months: number analyzed (Participants) | 14 | 16
  Role Functioning, Post-Treatment Follow Up 18 Months | 7.1 | 31.3
  Role Functioning, Post-Treatment Follow Up 24 Months: number analyzed (Participants) | 2 | 6
  Role Functioning, Post-Treatment Follow Up 24 Months | 0 | 16.7
  Social Functioning, Cycle 3 Day 1: number analyzed (Participants) | 455 | 442
  Social Functioning, Cycle 3 Day 1 | 29.0 | 31.2
  Social Functioning, Cycle 5 Day 1: number analyzed (Participants) | 439 | 422
  Social Functioning, Cycle 5 Day 1 | 29.6 | 30.6
  Social Functioning, Cycle 8 Day 1: number analyzed (Participants) | 413 | 403
  Social Functioning, Cycle 8 Day 1 | 21.8 | 25.8
  Social Functioning, Cycle 12 Day 1: number analyzed (Participants) | 376 | 357
  Social Functioning, Cycle 12 Day 1 | 18.9 | 19.0
  Social Functioning, Cycle 16 Day 1: number analyzed (Participants) | 333 | 312
  Social Functioning, Cycle 16 Day 1 | 19.5 | 17.6
  Social Functioning, Cycle 20 Day 1: number analyzed (Participants) | 252 | 234
  Social Functioning, Cycle 20 Day 1 | 20.2 | 16.2
  Social Functioning, Completion of Treatment/ Early Termination Visit: number analyzed (Participants) | 367 | 367
  Social Functioning, Completion of Treatment/ Early Termination Visit | 27.2 | 28.1
  Social Functioning, Post-Treatment Follow Up 3 Months: number analyzed (Participants) | 234 | 236
  Social Functioning, Post-Treatment Follow Up 3 Months | 26.5 | 25.4
  Social Functioning, Post-Treatment Follow Up 6 Months: number analyzed (Participants) | 148 | 164
  Social Functioning, Post-Treatment Follow Up 6 Months | 23.0 | 30.5
  Social Functioning, Post-Treatment Follow Up 9 Months: number analyzed (Participants) | 84 | 98
  Social Functioning, Post-Treatment Follow Up 9 Months | 22.6 | 32.7
  Social Functioning, Post-Treatment Follow Up 12 Months: number analyzed (Participants) | 45 | 58
  Social Functioning, Post-Treatment Follow Up 12 Months | 8.9 | 37.9
  Social Functioning, Post-Treatment Follow Up 18 Months: number analyzed (Participants) | 14 | 16
  Social Functioning, Post-Treatment Follow Up 18 Months | 14.3 | 37.5
  Social Functioning, Post-Treatment Follow Up 24 Months: number analyzed (Participants) | 2 | 6
  Social Functioning, Post-Treatment Follow Up 24 Months | 0 | 33.3
  Emotional Functioning, Cycle 3 Day 1: number analyzed (Participants) | 454 | 443
  Emotional Functioning, Cycle 3 Day 1 | 12.8 | 14.0
  Emotional Functioning, Cycle 5 Day 1: number analyzed (Participants) | 439 | 422
  Emotional Functioning, Cycle 5 Day 1 | 17.3 | 15.9
  Emotional Functioning, Cycle 8 Day 1: number analyzed (Participants) | 412 | 403
  Emotional Functioning, Cycle 8 Day 1 | 14.6 | 12.4
  Emotional Functioning, Cycle 12 Day 1: number analyzed (Participants) | 376 | 357
  Emotional Functioning, Cycle 12 Day 1 | 12.2 | 13.4
  Emotional Functioning, Cycle 16 Day 1: number analyzed (Participants) | 333 | 312
  Emotional Functioning, Cycle 16 Day 1 | 13.2 | 12.5
  Emotional Functioning, Cycle 20 Day 1: number analyzed (Participants) | 252 | 234
  Emotional Functioning, Cycle 20 Day 1 | 15.5 | 11.1
  Emotional Functioning, Completion of Treatment/ Early Termination Visit: number analyzed (Participants) | 368 | 367
  Emotional Functioning, Completion of Treatment/ Early Termination Visit | 19.3 | 19.3
  Emotional Functioning, Post-Treatment Follow Up 3 Months: number analyzed (Participants) | 234 | 236
  Emotional Functioning, Post-Treatment Follow Up 3 Months | 19.7 | 16.9
  Emotional Functioning, Post-Treatment Follow Up 6 Months: number analyzed (Participants) | 148 | 164
  Emotional Functioning, Post-Treatment Follow Up 6 Months | 20.9 | 14.6
  Emotional Functioning, Post-Treatment Follow Up 9 Months: number analyzed (Participants) | 84 | 98
  Emotional Functioning, Post-Treatment Follow Up 9 Months | 8.3 | 18.4
  Emotional Functioning, Post-Treatment Follow Up 12 Months: number analyzed (Participants) | 45 | 58
  Emotional Functioning, Post-Treatment Follow Up 12 Months | 8.9 | 22.4
  Emotional Functioning, Post-Treatment Follow Up 18 Months: number analyzed (Participants) | 14 | 16
  Emotional Functioning, Post-Treatment Follow Up 18 Months | 7.1 | 31.3
  Emotional Functioning, Post-Treatment Follow Up 24 Months: number analyzed (Participants) | 2 | 6
  Emotional Functioning, Post-Treatment Follow Up 24 Months | 0 | 66.7
  GHS/OoL Function, Cycle 3 Day 1: number analyzed (Participants) | 455 | 443
  GHS/OoL Function, Cycle 3 Day 1 | 24.2 | 22.8
  GHS/OoL Function, Cycle 5 Day 1: number analyzed (Participants) | 439 | 422
  GHS/OoL Function, Cycle 5 Day 1 | 24.1 | 23.7
  GHS/OoL Function, Cycle 8 Day 1: number analyzed (Participants) | 413 | 403
  GHS/OoL Function, Cycle 8 Day 1 | 21.3 | 18.1
  GHS/OoL Function, Cycle 12 Day 1: number analyzed (Participants) | 376 | 357
  GHS/OoL Function, Cycle 12 Day 1 | 17.6 | 13.2
  GHS/OoL Function, Cycle 16 Day 1: number analyzed (Participants) | 333 | 312
  GHS/OoL Function, Cycle 16 Day 1 | 18.3 | 13.5
  GHS/OoL Function, Cycle 20 Day 1: number analyzed (Participants) | 252 | 234
  GHS/OoL Function, Cycle 20 Day 1 | 20.2 | 11.1
  GHS/OoL Function, Completion of Treatment/ Early Termination Visit: number analyzed (Participants) | 368 | 367
  GHS/OoL Function, Completion of Treatment/ Early Termination Visit | 24.5 | 24.3
  GHS/OoL Function, Post-Treatment Follow Up 3 Months: number analyzed (Participants) | 234 | 236
  GHS/OoL Function, Post-Treatment Follow Up 3 Months | 20.5 | 22.9
  GHS/OoL Function, Post-Treatment Follow Up 6 Months: number analyzed (Participants) | 148 | 164
  GHS/OoL Function, Post-Treatment Follow Up 6 Months | 20.9 | 23.8
  GHS/OoL Function, Post-Treatment Follow Up 9 Months: number analyzed (Participants) | 84 | 98
  GHS/OoL Function, Post-Treatment Follow Up 9 Months | 21.4 | 25.5
  GHS/OoL Function, Post-Treatment Follow Up 12 Months: number analyzed (Participants) | 45 | 58
  GHS/OoL Function, Post-Treatment Follow Up 12 Months | 17.8 | 34.5
  GHS/OoL Function, Post-Treatment Follow Up 18 Months: number analyzed (Participants) | 14 | 16
  GHS/OoL Function, Post-Treatment Follow Up 18 Months | 21.4 | 43.8
  GHS/OoL Function, Post-Treatment Follow Up 24 Months: number analyzed (Participants) | 2 | 6
  GHS/OoL Function, Post-Treatment Follow Up 24 Months | 0 | 50.0
Statistical Analysis 1: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Emotional functioning, Cycle 3 Day 1; Test type: Superiority — Stratified Analysis; p = 0.6063, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.11, 95% CI 2-sided [0.75 to 1.63]
Statistical Analysis 2: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Emotional functioning, Cycle 5 Day 1; Test type: Superiority — Stratified Analysis; p = 0.5739, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.90, 95% CI 2-sided [0.63 to 1.29]
Statistical Analysis 3: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Emotional functioning, Cycle 8 Day 1; Test type: Superiority — Stratified Analysis; p = 0.3792, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.84, 95% CI 2-sided [0.56 to 1.25]
Statistical Analysis 4: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Emotional functioning, Cycle 12 Day 1; Test type: Superiority — Stratified Analysis; p = 0.6022, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.12, 95% CI 2-sided [0.73 to 1.73]
Statistical Analysis 5: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Emotional functioning, Cycle 16 Day 1; Test type: Superiority — Stratified Analysis; p = 0.7893, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.94, 95% CI 2-sided [0.59 to 1.49]
Statistical Analysis 6: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Emotional functioning, Cycle 20 Day 1; Test type: Superiority; p = 0.2125, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.71, 95% CI 2-sided [0.42 to 1.22]
Statistical Analysis 7: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Emotional functioning, Completion of Treatment/ Early Termination Visit; Test type: Superiority — Stratified Analysis; p = 0.9661, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.01, 95% CI 2-sided [0.70 to 1.46]
Statistical Analysis 8: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Emotional functioning, Post-Treatment Follow Up 3 Months; Test type: Superiority — Stratified Analysis; p = 0.4299, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.83, 95% CI 2-sided [0.52 to 1.32]
Statistical Analysis 9: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Emotional functioning, Post-Treatment Follow Up 6 Months; Test type: Superiority — Stratified Analysis; p = 0.1542, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.65, 95% CI 2-sided [0.36 to 1.18]
Statistical Analysis 10: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Emotional functioning, Post-Treatment Follow Up 9 Months; Test type: Superiority — Stratified Analysis; p = 0.0363, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 2.65, 95% CI 2-sided [1.04 to 6.76]
Statistical Analysis 11: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Emotional functioning, Post-Treatment Follow Up 12 Months; Test type: Superiority — Stratified Analysis; p = 0.0814, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 2.75, 95% CI 2-sided [0.85 to 8.93]
Statistical Analysis 12: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Emotional functioning, Post-Treatment Follow Up 18 Months; Test type: Superiority — Stratified Analysis; p = 0.1915, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 4.03, 95% CI 2-sided [0.43 to 38.00]
Statistical Analysis 13: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Emotional functioning, Post-Treatment Follow Up 24 Months; Test type: Superiority — Stratified Analysis; p = 0.3173, Cochran-Mantel-Haenszel; Difference in Proportion of Responders = 66.67, 95% CI 2-sided [-4.39 to 100.00]
Statistical Analysis 14: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Physical functioning, Cycle 3 Day 1; Test type: Superiority — Stratified Analysis; p = 0.9818, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.00, 95% CI 2-sided [0.73 to 1.35]
Statistical Analysis 15: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Physical functioning, Cycle 5 Day 1; Test type: Superiority — Stratified Analysis; p = 0.6263, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.08, 95% CI 2-sided [0.80 to 1.45]
Statistical Analysis 16: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Physical functioning, Cycle 8 Day 1; Test type: Superiority — Stratified Analysis; p = 0.9407, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.01, 95% CI 2-sided [0.73 to 1.40]
Statistical Analysis 17: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Physical functioning, Cycle 12 Day 1; Test type: Superiority — Stratified Analysis; p = 0.7700, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.94, 95% CI 2-sided [0.64 to 1.39]
Statistical Analysis 18: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Physical functioning, Cycle 16 Day 1; Test type: Superiority — Stratified Analysis; p = 0.8458, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.96, 95% CI 2-sided [0.63 to 1.45]
Statistical Analysis 19: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Physical functioning, Cycle 20 Day 1; Test type: Superiority — Stratified Analysis; p = 0.7028, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.91, 95% CI 2-sided [0.57 to 1.46]
Statistical Analysis 20: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Physical functioning, Completion of Treatment/ Early Termination Visit; Test type: Superiority; p = 0.1391, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.30, 95% CI 2-sided [0.92 to 1.83]
Statistical Analysis 21: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Physical functioning, Post-Treatment Follow Up 3 Months; Test type: Superiority — Stratified Analysis; p = 0.8002, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.06, 95% CI 2-sided [0.69 to 1.62]
Statistical Analysis 22: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Physical functioning, Post-Treatment Follow Up 6 Months; Test type: Superiority — Stratified Analysis; p = 0.9751, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.01, 95% CI 2-sided [0.60 to 1.68]
Statistical Analysis 23: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Physical functioning, Post-Treatment Follow Up 9 Months; Test type: Superiority — Stratified Analysis; p = 0.3811, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.37, 95% CI 2-sided [0.68 to 2.78]
Statistical Analysis 24: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Physical functioning, Post-Treatment Follow Up 12 Months; Test type: Superiority — Stratified Analysis; p = 0.3950, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.51, 95% CI 2-sided [0.58 to 3.90]
Statistical Analysis 25: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Physical functioning, Post-Treatment Follow Up 18 Months; Test type: Superiority — Stratified Analysis; p = 0.8993, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.89, 95% CI 2-sided [0.16 to 5.12]
Statistical Analysis 26: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Physical functioning, Post-Treatment Follow Up 24 Months; Test type: Superiority — Stratified; p = 0.3173, Cochran-Mantel-Haenszel; Difference in Proportion of Responders = 50.00, 95% CI 2-sided [-23.34 to 100.00]
Statistical Analysis 27: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Global health status/QoL, Cycle 3 Day 1; Test type: Superiority — Stratified Analysis; p = 0.5988, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.92, 95% CI 2-sided [0.68 to 1.25]
Statistical Analysis 28: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Global health status/QoL, Cycle 5 Day 1; Test type: Superiority — Stratified Analysis; p = 0.8859, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.98, 95% CI 2-sided [0.72 to 1.34]
Statistical Analysis 29: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Global health status/QoL, Cycle 8 Day 1; Test type: Superiority — Stratified Analysis; p = 0.2531, Cochran-Mantel-Haenszel; Stratified Analysis; Odds Ratio (OR) = 0.82, 95% CI 2-sided [0.58 to 1.16]
Statistical Analysis 30: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Global health status/QoL, Cycle 12 Day 1; Test type: Superiority — Stratified Analysis; p = 0.0785, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.69, 95% CI 2-sided [0.46 to 1.04]
Statistical Analysis 31: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Global health status/QoL, Cycle 16 Day 1; Test type: Superiority — Stratified Analysis; p = 0.0641, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.67, 95% CI 2-sided [0.43 to 1.03]
Statistical Analysis 32: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Global health status/QoL, Cycle 20 Day 1; Test type: Superiority — Stratified Analysis; p = 0.0046, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.48, 95% CI 2-sided [0.29 to 0.80]
Statistical Analysis 33: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Global health status/QoL, Completion of Treatment/ Early Termination Visit; Test type: Superiority — Stratified Analysis; p = 0.8928, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.98, 95% CI 2-sided [0.70 to 1.37]
Statistical Analysis 34: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Global health status/QoL, Post-Treatment Follow Up 3 Months; Test type: Superiority — Stratified Analysis; p = 0.6106, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.12, 95% CI 2-sided [0.72 to 1.74]
Statistical Analysis 35: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Global health status/QoL, Post-Treatment Follow Up 6 Months; Test type: Superiority — Stratified Analysis; p = 0.6159, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.15, 95% CI 2-sided [0.67 to 1.95]
Statistical Analysis 36: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Global health status/QoL, Post-Treatment Follow Up 9 Months; Test type: Superiority — Stratified Analysis; p = 0.5372, Cochran-Mantel-Haenszel; Stratified Analysis; Odds Ratio (OR) = 1.24, 95% CI 2-sided [0.62 to 2.49]
Statistical Analysis 37: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Global health status/QoL, Post-Treatment Follow Up 12 Months; Test type: Superiority — Stratified Analysis; p = 0.0845, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 2.22, 95% CI 2-sided [0.89 to 5.58]
Statistical Analysis 38: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Global health status/QoL, Post-Treatment Follow Up 18 Months; Test type: Superiority — Stratified Analysis; p = 0.1344, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 3.67, 95% CI 2-sided [0.62 to 21.56]
Statistical Analysis 39: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Global health status/QoL, Post-Treatment Follow Up 24 Months; Test type: Superiority — Stratified Analysis; p = 0.3173, Cochran-Mantel-Haenszel; Difference in Proportion of Responders = 50.00, 95% CI 2-sided [-23.34 to 100.00]
Statistical Analysis 40: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Role functioning, Cycle 3 Day 1; Test type: Superiority — Stratified Analysis; p = 0.0260, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.41, 95% CI 2-sided [1.04 to 1.92]
Statistical Analysis 41: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Role functioning, Cycle 5 Day 1; Test type: Superiority — Stratified Analysis; p = 0.9179, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.02, 95% CI 2-sided [0.75 to 1.37]
Statistical Analysis 42: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Role functioning, Cycle 8 Day 1; Test type: Superiority — Stratified Analysis; p = 0.5820, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.10, 95% CI 2-sided [0.79 to 1.53]
Statistical Analysis 43: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Role functioning, Cycle 12 Day 1; Test type: Superiority — Stratified Analysis; p = 0.9772, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.99, 95% CI 2-sided [0.67 to 1.47]
Statistical Analysis 44: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Role functioning, Cycle 16 Day 1; Test type: Superiority — Stratified Analysis; p = 0.1300, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.73, 95% CI 2-sided [0.49 to 1.10]
Statistical Analysis 45: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Role functioning, Cycle 20 Day 1; Test type: Superiority — Stratified Analysis; p = 0.0990, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.66, 95% CI 2-sided [0.40 to 1.08]
Statistical Analysis 46: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Role functioning, Completion of Treatment/ Early Termination Visit; Test type: Superiority — Stratified Analysis; p = 0.7133, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.07, 95% CI 2-sided [0.76 to 1.50]
Statistical Analysis 47: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Role functioning, Post-Treatment Follow Up 3 Months; Test type: Superiority — Stratified Analysis; p = 0.1384, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.38, 95% CI 2-sided [0.90 to 2.11]
Statistical Analysis 48: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Role functioning, Post-Treatment Follow Up 6 Months; Test type: Superiority — Stratified Analysis; p = 0.2895, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.33, 95% CI 2-sided [0.78 to 2.26]
Statistical Analysis 49: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Role functioning, Post-Treatment Follow Up 9 Months; Test type: Superiority — Stratified Analysis; p = 0.2221, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.55, 95% CI 2-sided [0.77 to 3.14]
Statistical Analysis 50: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Role functioning, Post-Treatment Follow Up 12 Months; Test type: Superiority — Stratified Analysis; p = 0.0005, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 7.37, 95% CI 2-sided [2.08 to 26.10]
Statistical Analysis 51: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Role functioning, Post-Treatment Follow Up 18 Months; Test type: Superiority; p = 0.2171, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 3.72, 95% CI 2-sided [0.40 to 34.56]
Statistical Analysis 52: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Role functioning, Post-Treatment Follow Up 24 Months; Test type: Superiority — Stratified Analysis; Difference in Proportion of Responders = 16.67, 95% CI 2-sided [-46.49 to 79.82]
Statistical Analysis 53: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Social functioning, Cycle 3 Day 1; Test type: Superiority — Stratified Analysis; p = 0.4647, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.11, 95% CI 2-sided [0.84 to 1.48]
Statistical Analysis 54: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Social functioning, Cycle 5 Day 1; Test type: Superiority — Stratified Analysis; p = 0.7676, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.04, 95% CI 2-sided [0.78 to 1.40]
Statistical Analysis 55: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Social functioning, Cycle 8 Day 1; Test type: Superiority — Stratified Analysis; p = 0.1983, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.24, 95% CI 2-sided [0.89 to 1.71]
Statistical Analysis 56: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Social functioning, Cycle 12 Day 1; Test type: Superiority — Stratified Analysis; p = 0.9874, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.00, 95% CI 2-sided [0.69 to 1.44]
Statistical Analysis 57: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Social functioning, Cycle 16 Day 1; Test type: Superiority — Stratified Analysis; p = 0.4716, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.86, 95% CI 2-sided [0.58 to 1.29]
Statistical Analysis 58: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Social functioning, Cycle 20 Day 1; Test type: Superiority — Stratified Analysis; p = 0.2041, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.74, 95% CI 2-sided [0.46 to 1.18]
Statistical Analysis 59: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Social functioning, Completion of Treatment/ Early Termination Visit; Test type: Superiority — Stratified Analysis; p = 0.7771, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.05, 95% CI 2-sided [0.76 to 1.45]
Statistical Analysis 60: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Social functioning, Post-Treatment Follow Up 3 Months; Test type: Superiority — Stratified Analysis; p = 0.8542, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.96, 95% CI 2-sided [0.64 to 1.45]
Statistical Analysis 61: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Social functioning, Post-Treatment Follow Up 6 Months; Test type: Superiority — Stratified Analysis; p = 0.1230, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.50, 95% CI 2-sided [0.90 to 2.50]
Statistical Analysis 62: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Social functioning, Post-Treatment Follow Up 9 Months; Test type: Superiority — Stratified Analysis; p = 0.1089, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.72, 95% CI 2-sided [0.88 to 3.34]
Statistical Analysis 63: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Social functioning, Post-Treatment Follow Up 12 Months; Test type: Superiority — Stratified Analysis; p = 0.0011, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 5.82, 95% CI 2-sided [1.85 to 18.30]
Statistical Analysis 64: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Social functioning, Post-Treatment Follow Up 18 Months; Test type: Superiority — Stratified Analysis; p = 0.2950, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 2.51, 95% CI 2-sided [0.43 to 14.74]
Statistical Analysis 65: Comparison: Placebo With Paclitaxel, Carboplatin and Bevacizumab vs Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Social functioning, Post-Treatment Follow Up 24 Months; Test type: Superiority — Stratified Analysis; Difference in Proportion of Responders = 33.33, 95% CI 2-sided [-37.72 to 100.00]

14. Secondary Outcome: Percentage of Participants With at Least One Adverse Event
Description: Percentage of participants with at least one adverse event.
Time Frame: From randomization up to approximately 59 months
Population: Safety-evaluable population is defined as patients who received any amount of any study treatment (atezolizumab, placebo, paclitaxel, carboplatin, or bevacizumab).
Measure: Number; unit: Percentage
Arm/Group | Placebo With Paclitaxel, Carboplatin and Bevacizumab | Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab
Number analyzed (Participants) | 644 | 642
Percentage | 99.8 | 100

15. Secondary Outcome: Maximum Serum Concentration (Cmax) of Atezolizumab
Time Frame: Cycle 1 Day 1 post dose and Cycle 3 Day 1 post dose
Population: PK-evaluable population is defined as patients who received any dose of study medication and who had at least one post-baseline PK sample available.
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab
Number analyzed (Participants) | 538
µg/mL
  Cycle 1 Day 1 | 487 (163)
  Cycle 3 Day 1: number analyzed (Participants) | 499
  Cycle 3 Day 1 | 614 (209)

16. Secondary Outcome: Minimum Serum Concentration (Cmin) of Atezolizumab
Time Frame: Cycle 2 Day 1 predose, Cycle 3 Day 1 Predose, Cycle 4 Day 1 predose, Cycle 8 Day 1 predose, Cycle 16 Day 1 predose
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab
Number analyzed (Participants) | 532
µg/mL
  Cycle 2 Day 1 | 88.9 (35.8)
  Cycle 3 Day 1: number analyzed (Participants) | 519
  Cycle 3 Day 1 | 146 (93.0)
  Cycle 4 Day 1: number analyzed (Participants) | 502
  Cycle 4 Day 1 | 149 (88.1)
  Cycle 8 Day 1: number analyzed (Participants) | 339
  Cycle 8 Day 1 | 242 (96.3)
  Cycle 16 Day 1: number analyzed (Participants) | 213
  Cycle 16 Day 1 | 286 (111)

17. Secondary Outcome: Percentage of Participants With Anti-Drug Antibodies (ADAs) to Atezolizumab
Time Frame: Baseline to approximately 55 months
Population: as for outcome 15
Measure: Number; unit: Percentage of participants
Arm/Group | Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab
Number analyzed (Participants) | 569
Percentage of participants
  Baseline evaluable participants: number analyzed (Participants) | 563
  Baseline evaluable participants | 0.7
  Post-baseline evaluable participants | 22.7

ADVERSE EVENTS:
Time Frame: From the first study drug to the data cutoff date: 12 August 2022 (up to 65 months)
Description: All-cause mortality reported for deaths that occurred during study based on ITT, which included all randomized participants. Serious & other adverse events reported based on safety population, which included participants who received any amount of any study drug.
Groups:
- Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab; Placebo With Paclitaxel, Carboplatin and Bevacizumab: Participants in the primary tumor-reductive surgery group received paclitaxel, carboplatin, atezolizumab placebo IV infusion on Day 1 of each 21-day cycle for a total of 6 cycles, and bevacizumab IV infusion starting with Cycle 2 for a total of 5 cycles, followed by maintenance therapy bevacizumab with atezolizumab placebo for a total of 22 cycles of atezolizumab placebo and 21 cycles of bevacizumab. Participants in the neoadjuvant therapy group received paclitaxel, carboplatin and placebo for 6 cycles and bevacizumab for 4 cycles. Interval surgery will occur between cycles 3 and 4. Each cycle is 21 days long. After 6 cycles, participants started maintenance therapy of bevacizumab and placebo for additional 16 cycles.
Arm/Group | Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab | Placebo With Paclitaxel, Carboplatin and Bevacizumab
All-Cause Mortality (participants affected / at risk) | 272/651 | 289/650
Serious Adverse Events (participants affected / at risk) | 304/642 | 215/644
Other Adverse Events (participants affected / at risk) | 637/642 | 637/644
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab (N=642) | Placebo With Paclitaxel, Carboplatin and Bevacizumab (N=644)
AGRANULOCYTOSIS (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
ANAEMIA (Blood and lymphatic system disorders) | 6 (7) | 10 (10)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 54 (59) | 24 (25)
GRANULOCYTOSIS (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
IMMUNE THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
LEUKOPENIA (Blood and lymphatic system disorders) | 3 (3) | 2 (2)
NEUTROPENIA (Blood and lymphatic system disorders) | 5 (5) | 5 (5)
PANCYTOPENIA (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 8 (11) | 10 (12)
THROMBOTIC MICROANGIOPATHY (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 2 (2) | 0 (0)
ANGINA UNSTABLE (Cardiac disorders) | 1 (1) | 0 (0)
ARRHYTHMIA (Cardiac disorders) | 1 (1) | 0 (0)
ATRIAL FIBRILLATION (Cardiac disorders) | 1 (1) | 0 (0)
ATRIAL TACHYCARDIA (Cardiac disorders) | 1 (1) | 0 (0)
ATRIAL THROMBOSIS (Cardiac disorders) | 1 (1) | 0 (0)
ATRIOVENTRICULAR BLOCK (Cardiac disorders) | 0 (0) | 1 (1)
CARDIAC ARREST (Cardiac disorders) | 2 (2) | 0 (0)
CARDIAC FAILURE (Cardiac disorders) | 1 (1) | 1 (1)
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 1 (1) | 0 (0)
CARDIOMYOPATHY (Cardiac disorders) | 1 (1) | 0 (0)
CARDIOVASCULAR DISORDER (Cardiac disorders) | 1 (1) | 0 (0)
MYOCARDIAL INFARCTION (Cardiac disorders) | 0 (0) | 1 (1)
MYOCARDIAL ISCHAEMIA (Cardiac disorders) | 1 (1) | 0 (0)
MYOCARDITIS (Cardiac disorders) | 0 (0) | 1 (1)
PALPITATIONS (Cardiac disorders) | 1 (1) | 0 (0)
OTOLITHIASIS (Ear and labyrinth disorders) | 0 (0) | 1 (1)
VERTIGO (Ear and labyrinth disorders) | 0 (0) | 3 (3)
ADDISON'S DISEASE (Endocrine disorders) | 1 (1) | 0 (0)
ADRENAL INSUFFICIENCY (Endocrine disorders) | 1 (1) | 0 (0)
AUTOIMMUNE THYROIDITIS (Endocrine disorders) | 1 (1) | 0 (0)
HYPERPARATHYROIDISM (Endocrine disorders) | 1 (1) | 0 (0)
HYPOTHYROIDISM (Endocrine disorders) | 2 (2) | 1 (1)
SECONDARY ADRENOCORTICAL INSUFFICIENCY (Endocrine disorders) | 1 (1) | 0 (0)
OCULAR MYASTHENIA (Eye disorders) | 1 (1) | 0 (0)
OPTIC NEUROPATHY (Eye disorders) | 1 (1) | 0 (0)
RETINAL VEIN OCCLUSION (Eye disorders) | 1 (1) | 0 (0)
ULCERATIVE KERATITIS (Eye disorders) | 1 (1) | 0 (0)
ABDOMINAL ADHESIONS (Gastrointestinal disorders) | 0 (0) | 1 (1)
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 0 (0) | 1 (1)
ABDOMINAL HERNIA (Gastrointestinal disorders) | 1 (1) | 0 (0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 9 (9) | 2 (2)
ABDOMINAL PAIN LOWER (Gastrointestinal disorders) | 0 (0) | 1 (1)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 (0) | 2 (2)
ANAL FISTULA (Gastrointestinal disorders) | 1 (1) | 0 (0)
ANAL HAEMORRHAGE (Gastrointestinal disorders) | 1 (2) | 0 (0)
ASCITES (Gastrointestinal disorders) | 0 (0) | 1 (1)
COLITIS (Gastrointestinal disorders) | 11 (12) | 6 (6)
CONSTIPATION (Gastrointestinal disorders) | 4 (4) | 5 (5)
DIARRHOEA (Gastrointestinal disorders) | 9 (11) | 11 (13)
DIARRHOEA HAEMORRHAGIC (Gastrointestinal disorders) | 1 (1) | 1 (1)
DIVERTICULAR PERFORATION (Gastrointestinal disorders) | 1 (1) | 0 (0)
DIVERTICULUM (Gastrointestinal disorders) | 0 (0) | 1 (1)
DUODENAL PERFORATION (Gastrointestinal disorders) | 0 (0) | 1 (1)
DYSPEPSIA (Gastrointestinal disorders) | 1 (1) | 0 (0)
DYSPHAGIA (Gastrointestinal disorders) | 1 (1) | 0 (0)
ENTERITIS (Gastrointestinal disorders) | 2 (2) | 0 (0)
ENTEROCOLITIS (Gastrointestinal disorders) | 1 (1) | 4 (4)
ENTEROCUTANEOUS FISTULA (Gastrointestinal disorders) | 0 (0) | 1 (1)
GASTRIC STENOSIS (Gastrointestinal disorders) | 1 (4) | 0 (0)
GASTRITIS (Gastrointestinal disorders) | 0 (0) | 1 (1)
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 1 (1)
GASTROINTESTINAL PERFORATION (Gastrointestinal disorders) | 2 (2) | 0 (0)
GINGIVAL PAIN (Gastrointestinal disorders) | 1 (1) | 0 (0)
HAEMORRHOIDAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 1 (1)
ILEAL PERFORATION (Gastrointestinal disorders) | 0 (0) | 1 (1)
ILEUS (Gastrointestinal disorders) | 12 (14) | 8 (10)
ILEUS PARALYTIC (Gastrointestinal disorders) | 0 (0) | 1 (1)
INCARCERATED INGUINAL HERNIA (Gastrointestinal disorders) | 0 (0) | 2 (2)
INCARCERATED UMBILICAL HERNIA (Gastrointestinal disorders) | 1 (1) | 0 (0)
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 8 (8) | 7 (9)
INTESTINAL PERFORATION (Gastrointestinal disorders) | 2 (2) | 3 (3)
LARGE INTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 1 (1)
LARGE INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 (1) | 2 (2)
LARGE INTESTINE PERFORATION (Gastrointestinal disorders) | 2 (2) | 0 (0)
LOWER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 2 (2) | 1 (1)
MECHANICAL ILEUS (Gastrointestinal disorders) | 0 (0) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 5 (5) | 5 (5)
OBSTRUCTION GASTRIC (Gastrointestinal disorders) | 1 (1) | 0 (0)
OESOPHAGITIS (Gastrointestinal disorders) | 1 (1) | 0 (0)
ORAL LICHEN PLANUS (Gastrointestinal disorders) | 1 (1) | 0 (0)
PANCREATIC FISTULA (Gastrointestinal disorders) | 2 (2) | 0 (0)
PANCREATITIS (Gastrointestinal disorders) | 1 (1) | 0 (0)
PERITONEAL ADHESIONS (Gastrointestinal disorders) | 1 (1) | 0 (0)
PNEUMATOSIS INTESTINALIS (Gastrointestinal disorders) | 0 (0) | 1 (1)
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 3 (3) | 1 (1)
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 10 (11) | 6 (6)
SMALL INTESTINAL PERFORATION (Gastrointestinal disorders) | 2 (2) | 0 (0)
SUBILEUS (Gastrointestinal disorders) | 0 (0) | 2 (2)
THROMBOSIS MESENTERIC VESSEL (Gastrointestinal disorders) | 1 (1) | 0 (0)
UMBILICAL HERNIA (Gastrointestinal disorders) | 1 (1) | 0 (0)
VOMITING (Gastrointestinal disorders) | 4 (5) | 7 (8)
ASTHENIA (General disorders) | 2 (2) | 0 (0)
CONDITION AGGRAVATED (General disorders) | 0 (0) | 1 (1)
DEATH (General disorders) | 2 (2) | 0 (0)
DEVICE RELATED THROMBOSIS (General disorders) | 1 (1) | 0 (0)
EARLY SATIETY (General disorders) | 1 (1) | 0 (0)
FATIGUE (General disorders) | 4 (4) | 2 (2)
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 3 (4) | 0 (0)
MUCOSAL INFLAMMATION (General disorders) | 1 (1) | 1 (1)
MULTIPLE ORGAN DYSFUNCTION SYNDROME (General disorders) | 0 (0) | 1 (1)
NON-CARDIAC CHEST PAIN (General disorders) | 2 (2) | 2 (2)
PAIN (General disorders) | 1 (1) | 0 (0)
PYREXIA (General disorders) | 26 (31) | 8 (9)
SYSTEMIC INFLAMMATORY RESPONSE SYNDROME (General disorders) | 1 (1) | 0 (0)
CHOLESTASIS (Hepatobiliary disorders) | 1 (1) | 0 (0)
DRUG-INDUCED LIVER INJURY (Hepatobiliary disorders) | 1 (1) | 0 (0)
HEPATIC FUNCTION ABNORMAL (Hepatobiliary disorders) | 1 (1) | 1 (1)
HEPATOTOXICITY (Hepatobiliary disorders) | 0 (0) | 2 (2)
IMMUNE-MEDIATED HEPATITIS (Hepatobiliary disorders) | 1 (1) | 0 (0)
JAUNDICE (Hepatobiliary disorders) | 0 (0) | 1 (1)
JAUNDICE CHOLESTATIC (Hepatobiliary disorders) | 1 (1) | 0 (0)
LIVER INJURY (Hepatobiliary disorders) | 4 (4) | 1 (1)
ANAPHYLACTIC REACTION (Immune system disorders) | 0 (0) | 2 (2)
ANAPHYLACTIC SHOCK (Immune system disorders) | 1 (1) | 1 (1)
CONTRAST MEDIA ALLERGY (Immune system disorders) | 1 (1) | 0 (0)
CYTOKINE RELEASE SYNDROME (Immune system disorders) | 1 (1) | 0 (0)
DRUG HYPERSENSITIVITY (Immune system disorders) | 1 (1) | 3 (3)
HYPERSENSITIVITY (Immune system disorders) | 0 (0) | 1 (1)
IMMUNE-MEDIATED ADVERSE REACTION (Immune system disorders) | 1 (1) | 0 (0)
SYSTEMIC IMMUNE ACTIVATION (Immune system disorders) | 2 (2) | 0 (0)
ABDOMINAL ABSCESS (Infections and infestations) | 5 (5) | 3 (3)
ABDOMINAL INFECTION (Infections and infestations) | 2 (2) | 0 (0)
APPENDICITIS (Infections and infestations) | 0 (0) | 2 (2)
BACTERAEMIA (Infections and infestations) | 0 (0) | 2 (3)
BRONCHITIS (Infections and infestations) | 2 (2) | 2 (2)
BRONCHITIS VIRAL (Infections and infestations) | 0 (0) | 1 (1)
CELLULITIS (Infections and infestations) | 3 (3) | 2 (2)
CLOSTRIDIUM DIFFICILE COLITIS (Infections and infestations) | 2 (2) | 0 (0)
CLOSTRIDIUM DIFFICILE INFECTION (Infections and infestations) | 1 (1) | 0 (0)
DEVICE RELATED INFECTION (Infections and infestations) | 1 (1) | 1 (1)
ENCEPHALITIS (Infections and infestations) | 1 (1) | 0 (0)
EPSTEIN-BARR VIRUS INFECTION (Infections and infestations) | 1 (1) | 0 (0)
ESCHERICHIA BACTERAEMIA (Infections and infestations) | 1 (1) | 0 (0)
FOURNIER'S GANGRENE (Infections and infestations) | 0 (0) | 1 (1)
GASTROENTERITIS CLOSTRIDIAL (Infections and infestations) | 1 (1) | 0 (0)
GINGIVITIS (Infections and infestations) | 1 (1) | 0 (0)
HERPES ZOSTER (Infections and infestations) | 0 (0) | 1 (1)
INFECTED LYMPHOCELE (Infections and infestations) | 4 (4) | 1 (1)
INFECTION (Infections and infestations) | 3 (3) | 1 (1)
INFECTIOUS MONONUCLEOSIS (Infections and infestations) | 1 (1) | 0 (0)
INFLUENZA (Infections and infestations) | 1 (1) | 1 (1)
KIDNEY INFECTION (Infections and infestations) | 0 (0) | 1 (1)
LYMPHANGITIS (Infections and infestations) | 0 (0) | 1 (1)
MENINGITIS BACTERIAL (Infections and infestations) | 1 (1) | 0 (0)
MENINGOENCEPHALITIS HERPETIC (Infections and infestations) | 1 (1) | 0 (0)
NASOPHARYNGITIS (Infections and infestations) | 0 (0) | 1 (1)
PELVIC ABSCESS (Infections and infestations) | 2 (2) | 1 (1)
PELVIC INFECTION (Infections and infestations) | 1 (1) | 1 (1)
PERITONITIS (Infections and infestations) | 4 (4) | 0 (0)
PERITONSILLITIS (Infections and infestations) | 0 (0) | 1 (1)
PNEUMONIA (Infections and infestations) | 10 (10) | 7 (7)
PNEUMONIA BACTERIAL (Infections and infestations) | 0 (0) | 1 (1)
PNEUMONIA VIRAL (Infections and infestations) | 0 (0) | 1 (1)
POSTOPERATIVE ABSCESS (Infections and infestations) | 1 (1) | 0 (0)
POSTOPERATIVE WOUND INFECTION (Infections and infestations) | 2 (2) | 0 (0)
PULPITIS DENTAL (Infections and infestations) | 0 (0) | 1 (1)
PYELONEPHRITIS (Infections and infestations) | 4 (5) | 3 (3)
PYELONEPHRITIS ACUTE (Infections and infestations) | 1 (1) | 0 (0)
SEPSIS (Infections and infestations) | 3 (3) | 9 (9)
SKIN INFECTION (Infections and infestations) | 1 (1) | 0 (0)
STAPHYLOCOCCAL SEPSIS (Infections and infestations) | 1 (1) | 0 (0)
TONSILLITIS (Infections and infestations) | 1 (1) | 0 (0)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 4 (4) | 1 (1)
URINARY TRACT INFECTION (Infections and infestations) | 9 (9) | 5 (6)
UROSEPSIS (Infections and infestations) | 4 (4) | 2 (2)
VAGINAL ABSCESS (Infections and infestations) | 1 (1) | 1 (1)
VAGINAL CELLULITIS (Infections and infestations) | 1 (1) | 0 (0)
VASCULAR DEVICE INFECTION (Infections and infestations) | 1 (1) | 1 (1)
WOUND INFECTION (Infections and infestations) | 0 (0) | 3 (3)
ANKLE FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
CONCUSSION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
FALL (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
FASCIAL RUPTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
FOOT FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
FRACTURED SACRUM (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
GASTROINTESTINAL ANASTOMOTIC LEAK (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
GASTROINTESTINAL INJURY (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
HIP FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
INCISION SITE IMPAIRED HEALING (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
INCISIONAL HERNIA (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
INFUSION RELATED REACTION (Injury, poisoning and procedural complications) | 5 (5) | 2 (2)
PERIPROSTHETIC FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
POST PROCEDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
PROCEDURAL INTESTINAL PERFORATION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
SPINAL COMPRESSION FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
VAGINAL CUFF DEHISCENCE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
WOUND COMPLICATION (Injury, poisoning and procedural complications) | 0 (0) | 2 (3)
WOUND DEHISCENCE (Injury, poisoning and procedural complications) | 2 (2) | 3 (5)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 1 (1) | 0 (0)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 1 (1) | 0 (0)
BLOOD CREATININE INCREASED (Investigations) | 1 (1) | 0 (0)
BLOOD POTASSIUM DECREASED (Investigations) | 1 (1) | 0 (0)
C-REACTIVE PROTEIN INCREASED (Investigations) | 1 (1) | 0 (0)
HEPATIC ENZYME INCREASED (Investigations) | 0 (0) | 2 (2)
INTERNATIONAL NORMALISED RATIO INCREASED (Investigations) | 1 (1) | 1 (1)
LIPASE INCREASED (Investigations) | 1 (1) | 0 (0)
LYMPHOCYTE COUNT DECREASED (Investigations) | 0 (0) | 1 (1)
NEUTROPHIL COUNT DECREASED (Investigations) | 3 (3) | 7 (7)
PLATELET COUNT DECREASED (Investigations) | 6 (9) | 10 (13)
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 3 (3) | 2 (3)
DECREASED APPETITE (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
DEHYDRATION (Metabolism and nutrition disorders) | 6 (6) | 0 (0)
ELECTROLYTE IMBALANCE (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
FOOD REFUSAL (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
HYPERCALCAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
HYPERMAGNESAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 4 (4) | 4 (5)
TYPE 1 DIABETES MELLITUS (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
MYALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
MYOPATHY (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
MYOSITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
SPINAL PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
ANAPLASTIC ASTROCYTOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
GASTROINTESTINAL STROMAL TUMOUR (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
INVASIVE DUCTAL BREAST CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
PAPILLARY THYROID CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
APHASIA (Nervous system disorders) | 1 (1) | 0 (0)
ATAXIA (Nervous system disorders) | 0 (0) | 1 (1)
CEREBELLAR INFARCTION (Nervous system disorders) | 0 (0) | 1 (1)
CEREBRAL INFARCTION (Nervous system disorders) | 1 (1) | 0 (0)
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 2 (3) | 3 (3)
COGNITIVE DISORDER (Nervous system disorders) | 1 (1) | 0 (0)
DEMENTIA (Nervous system disorders) | 1 (1) | 0 (0)
DEPRESSED LEVEL OF CONSCIOUSNESS (Nervous system disorders) | 0 (0) | 1 (1)
DIZZINESS (Nervous system disorders) | 0 (0) | 1 (1)
ENCEPHALOPATHY (Nervous system disorders) | 2 (2) | 0 (0)
EPILEPSY (Nervous system disorders) | 0 (0) | 1 (1)
HAEMORRHAGE INTRACRANIAL (Nervous system disorders) | 2 (2) | 1 (1)
HEADACHE (Nervous system disorders) | 0 (0) | 1 (1)
ISCHAEMIC STROKE (Nervous system disorders) | 1 (1) | 0 (0)
MYASTHENIA GRAVIS (Nervous system disorders) | 1 (1) | 0 (0)
NEUROPATHY PERIPHERAL (Nervous system disorders) | 1 (1) | 0 (0)
PERIPHERAL MOTOR NEUROPATHY (Nervous system disorders) | 1 (1) | 0 (0)
PRESYNCOPE (Nervous system disorders) | 2 (2) | 0 (0)
SEIZURE (Nervous system disorders) | 2 (3) | 0 (0)
SUBARACHNOID HAEMORRHAGE (Nervous system disorders) | 1 (1) | 1 (1)
SYNCOPE (Nervous system disorders) | 2 (2) | 2 (2)
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 4 (5) | 2 (2)
DELIRIUM (Psychiatric disorders) | 0 (0) | 1 (1)
DEPRESSION (Psychiatric disorders) | 1 (1) | 2 (3)
SUICIDAL IDEATION (Psychiatric disorders) | 0 (0) | 1 (1)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 3 (3) | 2 (2)
HAEMATURIA (Renal and urinary disorders) | 0 (0) | 1 (1)
HYDRONEPHROSIS (Renal and urinary disorders) | 1 (1) | 1 (1)
IMMUNE-MEDIATED NEPHRITIS (Renal and urinary disorders) | 0 (0) | 1 (1)
NEPHRITIS (Renal and urinary disorders) | 2 (2) | 0 (0)
NEPHROPATHY (Renal and urinary disorders) | 0 (0) | 1 (1)
PROTEINURIA (Renal and urinary disorders) | 3 (3) | 3 (3)
RENAL FAILURE (Renal and urinary disorders) | 1 (1) | 0 (0)
URINARY TRACT OBSTRUCTION (Renal and urinary disorders) | 0 (0) | 2 (2)
UROGENITAL FISTULA (Renal and urinary disorders) | 0 (0) | 1 (1)
FEMALE GENITAL TRACT FISTULA (Reproductive system and breast disorders) | 2 (2) | 2 (2)
VAGINAL FISTULA (Reproductive system and breast disorders) | 0 (0) | 1 (1)
ACUTE RESPIRATORY DISTRESS SYNDROME (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
HYPERVENTILATION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
LOWER RESPIRATORY TRACT CONGESTION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 2 (2)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 6 (6)
PULMONARY HAEMORRHAGE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
DRUG ERUPTION (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
DRUG REACTION WITH EOSINOPHILIA AND SYSTEMIC SYMPTOMS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
ECZEMA (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
ERYTHEMA MULTIFORME (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
LICHEN PLANUS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
RASH (Skin and subcutaneous tissue disorders) | 7 (7) | 0 (0)
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
SKIN ULCER (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
STEVENS-JOHNSON SYNDROME (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
TOXIC SKIN ERUPTION (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
URTICARIA (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
AORTIC DISSECTION (Vascular disorders) | 1 (1) | 0 (0)
CIRCULATORY COLLAPSE (Vascular disorders) | 1 (1) | 0 (0)
DEEP VEIN THROMBOSIS (Vascular disorders) | 2 (2) | 2 (2)
EMBOLISM (Vascular disorders) | 3 (3) | 3 (3)
EMBOLISM VENOUS (Vascular disorders) | 0 (0) | 2 (2)
HAEMORRHAGE (Vascular disorders) | 1 (1) | 0 (0)
HYPERTENSION (Vascular disorders) | 5 (5) | 4 (4)
HYPERTENSIVE URGENCY (Vascular disorders) | 1 (1) | 0 (0)
HYPOTENSION (Vascular disorders) | 1 (1) | 1 (1)
LYMPHOCELE (Vascular disorders) | 1 (1) | 2 (2)
LYMPHORRHOEA (Vascular disorders) | 0 (0) | 1 (1)
ORTHOSTATIC HYPOTENSION (Vascular disorders) | 1 (1) | 0 (0)
SHOCK HAEMORRHAGIC (Vascular disorders) | 1 (1) | 0 (0)
MYELOSUPPRESSION (Blood and lymphatic system disorders) | 3 (5) | 2 (2)
HEPATIC FAILURE (Hepatobiliary disorders) | 1 (1) | 0 (0)
SARCOIDOSIS (Immune system disorders) | 0 (0) | 1 (1)
BACTERIAL SEPSIS (Infections and infestations) | 1 (1) | 0 (0)
DIVERTICULITIS (Infections and infestations) | 0 (0) | 1 (1)
GASTROENTERITIS (Infections and infestations) | 1 (1) | 0 (0)
STOMA PROLAPSE (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
GLOMERULONEPHRITIS CHRONIC (Renal and urinary disorders) | 0 (0) | 1 (1)
HEAVY MENSTRUAL BLEEDING (Reproductive system and breast disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atezolizumab With Paclitaxel, Carboplatin and Bevacizumab (N=642) | Placebo With Paclitaxel, Carboplatin and Bevacizumab (N=644)
ANAEMIA (Blood and lymphatic system disorders) | 284 (468) | 266 (440)
LEUKOPENIA (Blood and lymphatic system disorders) | 69 (197) | 76 (243)
NEUTROPENIA (Blood and lymphatic system disorders) | 195 (477) | 197 (507)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 137 (278) | 134 (275)
HYPERTHYROIDISM (Endocrine disorders) | 51 (56) | 23 (26)
HYPOTHYROIDISM (Endocrine disorders) | 118 (131) | 54 (57)
VISION BLURRED (Eye disorders) | 31 (34) | 45 (48)
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 39 (51) | 49 (60)
ABDOMINAL PAIN (Gastrointestinal disorders) | 182 (253) | 173 (241)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 49 (56) | 66 (98)
CONSTIPATION (Gastrointestinal disorders) | 226 (297) | 240 (334)
DIARRHOEA (Gastrointestinal disorders) | 223 (336) | 199 (328)
DRY MOUTH (Gastrointestinal disorders) | 34 (39) | 18 (22)
DYSPEPSIA (Gastrointestinal disorders) | 44 (54) | 53 (61)
NAUSEA (Gastrointestinal disorders) | 325 (565) | 337 (628)
STOMATITIS (Gastrointestinal disorders) | 98 (138) | 67 (106)
VOMITING (Gastrointestinal disorders) | 150 (209) | 156 (230)
ASTHENIA (General disorders) | 78 (102) | 79 (117)
FATIGUE (General disorders) | 241 (297) | 251 (339)
MALAISE (General disorders) | 35 (59) | 33 (42)
MUCOSAL INFLAMMATION (General disorders) | 45 (49) | 26 (36)
OEDEMA PERIPHERAL (General disorders) | 40 (44) | 40 (42)
PYREXIA (General disorders) | 104 (124) | 54 (75)
NASOPHARYNGITIS (Infections and infestations) | 41 (60) | 41 (59)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 63 (83) | 55 (71)
URINARY TRACT INFECTION (Infections and infestations) | 109 (169) | 104 (140)
INFUSION RELATED REACTION (Injury, poisoning and procedural complications) | 78 (116) | 50 (71)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 91 (142) | 59 (100)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 89 (149) | 56 (93)
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 40 (50) | 33 (48)
LYMPHOCYTE COUNT DECREASED (Investigations) | 42 (55) | 24 (44)
NEUTROPHIL COUNT DECREASED (Investigations) | 177 (567) | 168 (610)
PLATELET COUNT DECREASED (Investigations) | 137 (267) | 142 (329)
WEIGHT DECREASED (Investigations) | 84 (91) | 68 (72)
WEIGHT INCREASED (Investigations) | 50 (51) | 44 (46)
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 143 (455) | 122 (535)
DECREASED APPETITE (Metabolism and nutrition disorders) | 119 (160) | 120 (154)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 46 (69) | 52 (85)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 72 (97) | 60 (94)
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 92 (134) | 83 (112)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 48 (63) | 45 (61)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 286 (444) | 285 (451)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 88 (97) | 90 (115)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 45 (70) | 51 (92)
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 45 (50) | 44 (57)
MYALGIA (Musculoskeletal and connective tissue disorders) | 144 (205) | 163 (239)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 34 (34) | 32 (35)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 81 (110) | 89 (121)
DIZZINESS (Nervous system disorders) | 76 (93) | 80 (102)
DYSGEUSIA (Nervous system disorders) | 56 (66) | 50 (52)
HEADACHE (Nervous system disorders) | 149 (220) | 179 (278)
HYPOAESTHESIA (Nervous system disorders) | 50 (63) | 59 (78)
NEUROPATHY PERIPHERAL (Nervous system disorders) | 152 (175) | 166 (196)
PARAESTHESIA (Nervous system disorders) | 47 (57) | 40 (65)
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 178 (201) | 163 (186)
ANXIETY (Psychiatric disorders) | 38 (43) | 49 (58)
DEPRESSION (Psychiatric disorders) | 35 (41) | 38 (41)
INSOMNIA (Psychiatric disorders) | 89 (100) | 97 (119)
PROTEINURIA (Renal and urinary disorders) | 137 (172) | 140 (178)
COUGH (Respiratory, thoracic and mediastinal disorders) | 102 (127) | 80 (101)
DYSPHONIA (Respiratory, thoracic and mediastinal disorders) | 44 (47) | 44 (50)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 87 (112) | 86 (110)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 136 (166) | 139 (178)
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 32 (38) | 36 (40)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 47 (58) | 41 (50)
ALOPECIA (Skin and subcutaneous tissue disorders) | 386 (393) | 410 (415)
DRY SKIN (Skin and subcutaneous tissue disorders) | 35 (37) | 33 (39)
PRURITUS (Skin and subcutaneous tissue disorders) | 87 (108) | 61 (74)
RASH (Skin and subcutaneous tissue disorders) | 152 (205) | 99 (119)
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 45 (67) | 17 (19)
URTICARIA (Skin and subcutaneous tissue disorders) | 33 (49) | 10 (12)
HOT FLUSH (Vascular disorders) | 35 (37) | 48 (57)
HYPERTENSION (Vascular disorders) | 225 (354) | 263 (392)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 28 (29) | 33 (39)
PAIN (General disorders) | 33 (35) | 32 (39)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2021-11-22): https://cdn.clinicaltrials.gov/large-docs/00/NCT03038100/Prot_000.pdf
  • Statistical Analysis Plan (2021-12-06): https://cdn.clinicaltrials.gov/large-docs/00/NCT03038100/SAP_001.pdf